CLINICAL TRIAL: NCT00310375
Title: A Multicenter, Open-label, Long-term, Safety, Tolerability and Efficacy Study of Retigabine in Adult Epilepsy Patients With Partial-onset Seizures (Extension of Study VRX-RET-E22-301)
Brief Title: Open-label Extension Study of the Phase 3 VRX-RET-E22-301 Double-Blind Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VRX-RET-E22-303; RTG115098 (Other: GlaxoSmithKline)
Record Dates: First submitted 2006-03-30; First posted 2006-04-03 (Estimated); Results first posted 2016-11-25 (Estimated); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Epilepsy
Keywords: Epilepsy; Partial Seizures; Potassium Channels; Anticonvulsant; Complex Partial Seizures; Epilepsies, Partial; RTG115098
MeSH Terms: conditions — Epilepsy; Seizures; Epilepsies, Partial | interventions — ezogabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ezogabine: USAN Retigabine (International Nonproprietary Name) (Experimental): Film-coated tablets - 50mg, 100mg or 300mg
  Interventions: Drug: Ezogabine: USAN Retigabine (International Nonproprietary Name)

INTERVENTIONS:
Drug: Ezogabine: USAN Retigabine (International Nonproprietary Name) — Film-coated tablets containing 50 mg, 100 mg, or 300 mg of retigabine per tablet. Dosage and frequency will be specific to each patient so long as the patient receives between 600 and 1200 mg of retigabine per day. The duration will be until the trial concludes or the patient leaves the trial.
  Other Names: GKE-841; D-23129; GW582892X

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of long-term therapy with retigabine administered as adjunctive therapy in adult epilepsy patients with partial-onset seizures, who completed the VRX-RET-E22-301 double-blind study. The efficacy of long-term treatment with retigabine and patient quality of life will also be assessed.

DETAILED DESCRIPTION:
This Phase 3 trial is an open-label extension study of the placebo-controlled, double-blind VRX-RET-E22-301 trial. Patients who have completed the VRX-RET-E22-301 trial and who meet inclusion and exclusion criteria will be treated with 600-1200 mg/day of retigabine as an adjunct therapy to their current antiepileptic drugs (AEDs) or vagal nerve stimulation. Treatment will be continued until retigabine is commercially available, or until the program is discontinued. Patients will be recruited from 45-50 sites in the United States, Canada, Mexico, Brazil, and Argentina. The safety and tolerability of long-term therapy with retigabine administered as adjunctive therapy in adult epilepsy patients with partial-onset seizures will be evaluated. In addition, the efficacy of long-term treatment with retigabine and patient quality of life will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patient has successfully completed the Maintenance and Transition phases of Study VRX-RET-E22-301 for the treatment of partial-onset seizures
* Patient is expected to benefit from participation in the study in the opinion of the Investigator.

Exclusion Criteria:

* Patient meets any of the withdrawal criteria in the previous VRX-RET-E22-301 study or is experiencing an ongoing serious adverse event.
* Patient is receiving any investigational drug or using any experimental device in addition to Retigabine for treatment of epilepsy or any other medical condition.
* Patient has any other condition that would prevent compliance with the study procedures or proper reporting of adverse events.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2006-05-01 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2017-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (51):
- United States (30):
  - University of Alabama -- Department of Neurology/Epilepsy Center, Birmingham, Alabama
  - North Alabama Neuroscience Research Associates, Huntsville, Alabama
  - Neurology Clinic, Northport, Alabama
  - Barrow Neurological Institute, Phoenix, Arizona
  - Clinical Trials Inc., Little Rock, Arkansas
  - UCSD Thornton Hospital, La Jolla, California
  - University of Southern California -- Keck School of Medicine, Los Angeles, California
  - West Los Angeles VA Healthcare Center, Los Angeles, California
  - Delta Waves, Colorado Springs, Colorado
  - University of Colorado Department Of Neurology, Denver, Colorado
  - University of Florida -- Shands Jacksonville, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Lovelace Scientific Resources, Sarasota, Florida
  - McFarland Clinic, Ames, Iowa
  - University of Kentucky, Lexington, Kentucky
  - Mid-Atlantic Epilepsy and Sleep Center, Bethesda, Maryland
  - Henry Ford Hospital, Detroit, Michigan
  - Minnesota Epilepsy Group, P.A., Saint Paul, Minnesota
  - The Comprehensive Epilepsy Care Center for Children and Adults, Chesterfield, Missouri
  - Beth Israel Medical Center, New York, New York
  - Asheville Neurology Specialists, Asheville, North Carolina
  - Medical University of Ohio at Toledo, Toledo, Ohio
  - Oregon Neurology PC, Tualatin, Oregon
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Medical City Dallas Hospital, Dallas, Texas
  - Neurological Clinic of Texas, Dallas, Texas
  - Memorial Hermann Hospital, Houston, Texas
  - University of Virginia Comprehensive Epilepsy Program, Charlottesville, Virginia
  - Virginia Commonwealth University Medical Center, Richmond, Virginia
- Argentina (6):
  - Hospital Italiano de Buenos Aires, Capital Federal, CBA
  - Hospital General de Agudos "Dr. J.M. Ramos Mejia", Capital Federal, CBA
  - Hospital General de Agudos "Dr. Teodoro Alvarez", Capital Federal, CBA
  - Fundacion Lennox, Córdoba, CRD
  - Sanatorio del Salvador II, Córdoba, CRD
  - Hospital Privado Centro Medico de Cordoba, Córdoba, CRD
- Brazil (4):
  - Hospital Universitario Prof Edgard Santos -- UFBA, Salvador, Estado de Bahia
  - Hospital das Clinicas de Ribeirao Preto -- Universidade de Sa Neurologia, Ribeirão Preto, São Paulo
  - Hospital Sao Paulo -- Escola Paulista de Medicina -- UNIFESP, São Paulo, São Paulo
  - Hospital das Clinicas da Fac de Medicina de Sao Paulo, São Paulo, São Paulo
- Canada (4):
  - Foothills Medical Center, Calgary, Alberta
  - Glenrose Rehabilitation Center, Edmonton, Alberta
  - Health Sciences Centre, St. John's, Newfoundland and Labrador
  - CHUM -- Hôpital Notre-Dame, Montreal, Quebec
- Mexico (7):
  - Antiguo Hospital Civil de Guadalajara, Guadalajara, Jalisco
  - Instituto Nacional de Neurologia y Neurocirugia, La Fama, Mexico City
  - Centro Medico, Mexico City, Mexico City
  - Hospital de Psiquiatria San Fernando, IMSS, Mexico City, Mexico City
  - CIF BIOTEC, Medica Sur, Tlalpan, Mexico City
  - Hospital y Clinica OCA S.A. de C.V., Monterrey, Nuevo León
  - Hospital Central Dr. Ignacio Morones Prieto, San Luis Potosí City, San Luis Potosí

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20375

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible Participants (Par) who completed the Maintenance and Transition Phases of the parent study were enrolled in this open-label extension study. Par received 600-1200 mg/day retigabine as an adjunct therapy to current antiepileptic medication or vagal nerve stimulation until Par was withdrawn or withdrew consent or until study was terminated.
Pre-assignment Details: All participants who completed Study VRX-RET-E22-301(parent study) and did not have an ongoing serious adverse event (SAE) were eligible to participate in the study.
Groups:
- Placebo in Parent Study: Participants received retigabine tablets as a total dose of between 600 to 1200 mg/day (dose administered twice daily or TID) as an adjunct therapy to their ongoing antiepileptic drugs with or without vagal nerve stimulation until withdrawal, withdrawn consent or switched to commercial product. Participants who received placebo in parent study are included in this arm.
- Retigabine in Parent Study: Participants received retigabine tablets as a total dose of between 600 to 1200 mg/day (dose administered twice daily or TID) as an adjunct therapy to their ongoing antiepileptic drugs with or without vagal nerve stimulation until withdrawal, withdrawn consent or switched to commercial product. Participants who received retigabine in parent study are included in this arm.
- Safety Follow-up Continuation Phase (SFUCP): Participants who withdraw from retigabine and who were found to have abnormal pigmentation of the retina or unexplained vision loss, pigmentation of non-retinal ocular tissue or discoloration of skin, lips, nails or mucosa entered the SFUCP. During the SFUCP, participants underwent 6-monthly comprehensive eye examinations and/or skin assessments by the investigator, ophthalmologist, retinal specialist or dermatologist as appropriate. Participants were followed up in the SFUCP until the dermatology/ophthalmology finding(s) either resolved or stabilized. Stabilization was defined in the protocol as no changes on two consecutive 6-monthly assessments over at least over 12 months after discontinuation of retigabine.
Period: Primary Reporting Phase
Arm/Group | Placebo in Parent Study | Retigabine in Parent Study | Safety Follow-up Continuation Phase (SFUCP)
Started | 102 | 79 | 0
Completed | 11 | 11 | 0
Not Completed | 91 | 68 | 0
Not completed — Adverse Event | 28 | 22 | 0
Not completed — Lack of Efficacy | 24 | 19 | 0
Not completed — Pregnancy | 2 | 2 | 0
Not completed — Withdrawal by Subject | 10 | 7 | 0
Not completed — Protocol Violation | 8 | 5 | 0
Not completed — Change in Par medical condition | 2 | 0 | 0
Not completed — Transaminase >5 upper limit of normal | 2 | 1 | 0
Not completed — Physician Decision | 5 | 3 | 0
Not completed — Request of the sponsor | 2 | 2 | 0
Not completed — Failed to return | 1 | 3 | 0
Not completed — Participant request unrelated to study | 1 | 2 | 0
Not completed — Going for temporal lobectomy | 1 | 0 | 0
Not completed — Missed study drug >5 days | 1 | 0 | 0
Not completed — Site closure | 3 | 0 | 0
Not completed — Missed study drug for 2 months | 1 | 0 | 0
Not completed — Par. switched to commercial product | 0 | 1 | 0
Not completed — Request of Ethics Committee | 0 | 1 | 0
Period: Safety Follow-up Continuation Phase
Arm/Group | Placebo in Parent Study | Retigabine in Parent Study | Safety Follow-up Continuation Phase (SFUCP)
Started | 0 | 0 | 19
Completed | 0 | 0 | 18 (Met the protocol defined stopping criteria)
Not Completed | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo in Parent Study | Retigabine in Parent Study | Total
Number analyzed (Participants) | 102 | 79 | 181
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.0 (11.74) | 37.1 (12.20) | 37.6 (11.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 39 | 94
  Male | 47 | 40 | 87
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 54 | 40 | 94
  Hispanic | 30 | 26 | 56
  African-American (black) | 7 | 7 | 14
  Other | 11 | 6 | 17
Number of Participants with Vagal nerve stimulator (VNS) use [Number; unit: Participants]
  No | 89 | 74 | 163
  Yes | 13 | 5 | 18
Number of background AEDs [Number; unit: Participants]
  AED=1 | 12 | 18 | 30
  AED=2 | 47 | 41 | 88
  AED=3 | 43 | 20 | 63
Mean Duration of Partial seizures [Mean (Standard Deviation); unit: Years] — For this study specific outcome measure, Placebo in Parent Study N=101 and Retigabine in parent study N=79
  Years | 24.1 (13.06) | 23.7 (12.88) | 23.9 (12.95)
Mean Duration of Generalized Seizure [Mean (Standard Deviation); unit: Years] — For this study specific outcome measure, Placebo in Parent Study N=12 and Retigabine in parent study N=8
  Years | 18.6 (12.45) | 25.8 (13.25) | 21.5 (12.94)
Clinical Global Impression (CGI) at Baseline [Number; unit: Participants]
  Not Assessed | 0 | 0 | 0
  No Seizures | 0 | 0 | 0
  Very Mild Severity | 2 | 0 | 2
  Mild Severity | 9 | 8 | 17
  Moderate Severity | 49 | 40 | 89
  Marked Severity | 36 | 26 | 62
  Very Severe | 6 | 5 | 11
  Among the Most Extremely Severe | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Serious Adverse Event (SAE) and Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization (unplanned hospital stay) or prolongation of existing hospitalization, results in disability/incapacity or is a congenital anomaly/birth defect. Treatment-emergent AE was defined as an AE with an onset on or after the day of first dose of the study medication and on or before 30 days after the last dose date. AEs reported during parent study and worsened after first dose of RTG in this OLE study were also reported.
Time Frame: Assessed up to a maximum of 9 years
Population: Safety Population included all participants who took at least 1 dose of study medication
Measure: Number; unit: Participants
Groups:
- Overall Study: Participants received retigabine tablets for a total dose of between 600 to 1200 mg/day (dose administered twice daily or TID) as an adjunct therapy to their ongoing antiepileptic drugs with or without vagal nerve stimulation treatment until withdrawal, withdrawn consent or switched to commercial product.
Arm/Group | Overall Study
Number analyzed (Participants) | 181
Participants
  Any Treatment-emergent SAE | 48
  Any Treatment-emergent AE | 173

2. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events Leading to Withdrawal From Study Drug
Description: Treatment-emergent AE was defined as an AE with an onset on or after the day of first dose of the study medication and on or before 30 days after the last dose date. AEs reported during parent study and worsened after first dose of RTG in this OLE study were also reported.
Time Frame: Assessed up to a maximum of 9 years
Population: Safety Population
Measure: Number; unit: Participants.
Arm/Group | Overall Study
Number analyzed (Participants) | 181
Participants. | 52

3. Primary Outcome: Kaplan-Meier Estimate of the Probability of Discontinuation (d/c) From Study Drug
Description: The time frame of premature study discontinuation was defined as the time from the day of first the study medication to the time of withdrawal from study drug. For those who have a taper dose start date, the time of withdrawal was the day before the start of taper dose. For those without a taper dose start date, the time of withdrawal was the last dose date. Participants who switched to the commercial product were censored at the last dose of study drug in the Kaplan-Meier analysis. All participants who withdrew from study drug prematurely but didn't switch to commercial product were counted as "events". Kaplan-Meier estimate of the probability of discontinuation at the specified time or earlier. Number of Participants continuing on RTG at each time of withdrawal were analyzed (represented as n=X in category title).
Time Frame: Assessed up to a maximum of 9 years
Population: Safety Population
Measure: Number; unit: Percentage Probability of d/c
Arm/Group | Overall Study
Number analyzed (Participants) | 181
Percentage Probability of d/c
  Day 0,n= 181 | 0.0
  Day 2,n= 180 | 0.6
  Day 6,n= 179 | 1.1
  Day 8,n= 178 | 1.7
  Day 12,n= 177 | 2.2
  Day 13,n= 176 | 2.8
  Day 18,n= 175 | 3.3
  Day 20,n= 174 | 3.9
  Day 21,n= 173 | 4.4
  Day 26,n= 172 | 5.0
  Day 27,n= 170 | 6.1
  Day 28,n= 169 | 6.6
  Day 29,n= 168 | 7.2
  Day 30,n= 167 | 7.7
  Day 32,n= 166 | 8.3
  Day 33,n= 164 | 9.4
  Day 39,n= 163 | 9.9
  Day 50,n= 162 | 10.5
  Day 52,n= 161 | 11.0
  Day 55,n= 160 | 11.6
  Day 67,n= 158 | 12.7
  Day 85,n= 157 | 13.3
  Day 89,n= 155 | 14.4
  Day 91,n= 153 | 15.5
  Day 93,n= 152 | 16.0
  Day 96,n= 151 | 16.6
  Day 109,n= 150 | 17.1
  Day 118,n= 149 | 17.7
  Day 119,n= 148 | 18.2
  Day 124,n= 147 | 18.8
  Day 134,n= 146 | 19.3
  Day 135,n= 145 | 19.9
  Day 140,n= 144 | 20.4
  Day 144,n= 143 | 21.0
  Day 166,n= 142 | 21.5
  Day 167,n= 141 | 22.1
  Day 175,n= 140 | 22.7
  Day 179,n= 139 | 23.2
  Day 180,n= 138 | 23.8
  Day 181,n= 137 | 24.3
  Day 182,n= 135 | 25.4
  Day 185,n= 134 | 26.0
  Day 188,n= 133 | 26.5
  Day 207,n= 132 | 27.1
  Day 210,n= 131 | 27.6
  Day 211,n= 130 | 28.2
  Day 213,n= 129 | 28.7
  Day 216,n= 128 | 29.3
  Day 224,n= 127 | 29.8
  Day 231,n= 126 | 30.4
  Day 237,n= 125 | 30.9
  Day 240,n= 124 | 31.5
  Day 253,n= 123 | 32.0
  Day 271,n= 122 | 32.6
  Day 278,n= 121 | 33.1
  Day 280,n= 120 | 33.7
  Day 281,n= 119 | 34.3
  Day 282,n= 118 | 34.8
  Day 303,n= 117 | 35.4
  Day 315,n= 116 | 35.9
  Day 336,n= 114 | 37.0
  Day 338,n= 113 | 37.6
  Day 358,n= 112 | 38.1
  Day 361,n= 111 | 38.7
  Day 362,n= 110 | 39.2
  Day 372,n= 109 | 39.8
  Day 377,n= 108 | 40.3
  Day 392,n= 107 | 40.9
  Day 407,n= 106 | 41.4
  Day 413,n= 105 | 42.0
  Day 477,n= 104 | 42.5
  Day 479,n= 103 | 43.1
  Day 483,n= 102 | 43.6
  Day 489,n= 101 | 44.2
  Day 535,n= 100 | 44.8
  Day 593,n= 99 | 45.3
  Day 602,n= 98 | 45.9
  Day 603,n= 97 | 46.4
  Day 606,n= 96 | 47.0
  Day 609,n= 95 | 47.5
  Day 660,n= 94 | 48.1
  Day 685,n= 93 | 48.6
  Day 722,n= 92 | 49.2
  Day 783,n= 91 | 49.7
  Day 821,n= 90 | 50.3
  Day 843,n= 88 | 51.4
  Day 848,n= 87 | 51.9
  Day 881,n= 86 | 52.5
  Day 959,n= 85 | 53.0
  Day 1076,n= 84 | 53.6
  Day 1080,n= 83 | 54.1
  Day 1084,n= 82 | 54.7
  Day 1090,n= 81 | 55.2
  Day 1119,n= 80 | 55.8
  Day 1146,n= 79 | 56.4
  Day 1196,n= 78 | 56.9
  Day 1210,n= 77 | 57.5
  Day 1225,n= 76 | 58.0
  Day 1322,n= 75 | 58.6
  Day 1326,n= 74 | 59.1
  Day 1338,n= 73 | 59.7
  Day 1339,n= 72 | 60.2
  Day 1407,n= 71 | 60.8
  Day 1429,n= 70 | 61.3
  Day 1520,n= 69 | 61.9
  Day 1561,n= 68 | 62.4
  Day 1563,n= 67 | 63.0
  Day 1619,n= 66 | 63.0
  Day 1645,n= 65 | 63.0
  Day 1655,n= 64 | 63.0
  Day 1656,n= 63 | 63.0
  Day 1673,n= 62 | 63.6
  Day 1676,n= 61 | 64.2
  Day 1686,n= 60 | 64.7
  Day 1737,n= 59 | 64.7
  Day 1780,n= 58 | 64.7
  Day 1800,n= 57 | 65.4
  Day 1811,n= 56 | 66.0
  Day 1813,n= 55 | 66.6
  Day 1862,n= 54 | 66.6
  Day 1885,n= 53 | 67.2
  Day 1911,n= 52 | 67.2
  Day 1926,n= 51 | 67.2
  Day 1933,n= 50 | 67.2
  Day 1952,n= 49 | 67.8
  Day 1989,n= 48 | 67.8
  Day 1994,n= 47 | 68.5
  Day 2008,n= 46 | 68.5
  Day 2038,n= 45 | 68.5
  Day 2044,n= 44 | 69.2
  Day 2051,n= 43 | 69.9
  Day 2073,n= 42 | 69.9
  Day 2109,n= 41 | 69.9
  Day 2111,n= 40 | 69.9
  Day 2139,n= 39 | 69.9
  Day 2157,n= 38 | 69.9
  Day 2161,n= 37 | 70.7
  Day 2164,n= 36 | 71.5
  Day 2170,n= 35 | 72.3
  Day 2228,n= 34 | 72.3
  Day 2234,n= 33 | 72.3
  Day 2248,n= 32 | 72.3
  Day 2274,n= 31 | 73.2
  Day 2278,n= 30 | 73.2
  Day 2282,n= 28 | 74.9
  Day 2290,n= 27 | 75.8
  Day 2294,n= 26 | 76.7
  Day 2297,n= 25 | 77.6
  Day 2301,n= 24 | 78.5
  Day 2337,n= 23 | 79.4
  Day 2393,n= 22 | 80.3
  Day 2523,n= 21 | 81.2
  Day 2527,n= 20 | 82.1
  Day 2528,n= 19 | 83.0
  Day 2535,n= 18 | 83.9
  Day 2646,n= 16 | 85.7
  Day 2702,n= 15 | 86.6
  Day 2735,n= 14 | 87.5
  Day 2768,n= 13 | 88.4
  Day 2792,n= 12 | 89.3
  Day 2795,n= 11 | 90.2
  Day 2833,n= 10 | 91.1
  Day 2848,n= 9 | 91.9
  Day 2871,n= 8 | 92.8
  Day 2886,n= 7 | 93.7
  Day 3001,n= 6 | 94.6
  Day 3004,n= 5 | 95.5
  Day 3023,n= 4 | 96.4
  Day 3091,n= 3 | 97.3
  Day 3092,n= 2 | 98.2
  Day 3101,n= 1 | 99.1
  Day 3186,n= 0 | 100.0

4. Primary Outcome: Change From Baseline in Blood Pressure
Description: Systolic blood pressure (SBP) and diastolic blood pressure (DBP) was obtained in supine (Su) position and again in standing (St) position after the participant was standing for approximately 2 minutes at each study visit (Month 1, Month 3, Month 6, Month 9, Month 12 and every 4 months after Month 12). Baseline assessment in this study is defined as the last assessment for the endpoint in parent study taken prior to the first active treatment with Retigabine. Change from Baseline was calculated as post-Baseline value minus Baseline value. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles). Not Applicable (NA) indicates that data were not available.
Time Frame: Baseline and Up to Month 108
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimeter of mercury (mmHg)
Arm/Group | Overall Study
Number analyzed (Participants) | 181
Millimeter of mercury (mmHg)
  Su DBP Mon 1, n=173 | -1.1 (9.74)
  Su DBP Mon 3, n=159 | -0.7 (9.73)
  Su DBP Mon 6, n=143 | -2.9 (10.61)
  Su DBP Mon 9, n=125 | -2.6 (10.72)
  Su DBP Mon 12, n=173 | -0.6 (11.08)
  Su DBP Mon 16, n=104 | -2.3 (11.69)
  Su DBP Mon 20, n=100 | -1.9 (13.12)
  Su DBP Mon 24, n=112 | -1.3 (11.24)
  Su DBP Mon 28, n=88 | -0.8 (12.75)
  Su DBP Mon 32, n=85 | -0.6 (11.18)
  Su DBP Mon 36, n=92 | -1.6 (10.81)
  Su DBP Mon 40, n=78 | -2.5 (11.62)
  Su DBP Mon 44, n=76 | -1.1 (11.75)
  Su DBP Mon 48, n=82 | -1.2 (11.76)
  Su DBP Mon 52, n=68 | 0.7 (9.74)
  Su DBP Mon 56, n=63 | -0.3 (11.37)
  Su DBP Mon 60, n=70 | -0.8 (11.67)
  Su DBP Mon 64, n=50 | -1.7 (11.34)
  Su DBP Mon 68, n=45 | -1.1 (11.24)
  Su DBP Mon 72, n=57 | 0.2 (11.02)
  Su DBP Mon 76, n=31 | -0.5 (9.01)
  Su DBP Mon 80, n=24 | -1 (7.13)
  Su DBP Mon 84, n=36 | -2.3 (11.04)
  Su DBP Mon 88, n=17 | -0.1 (6.94)
  Su DBP Mon 92, n=16 | -2.8 (8.49)
  Su DBP Mon 96, n=19 | -0.2 (8.3)
  Su DBP Mon 100, n=7 | -6.3 (3.25)
  Su DBP Mon 104, n=1 | -20.0 (NA) — Standard deviation value was not available as only one participant was analyzed
  Su DBP Mon 108, n=10 | -2.0 (7.27)
  St DBP Mon 1, n=173 | -0.5 (9.97)
  St DBP Mon 3, n=159 | -1.0 (11.68)
  St DBP Mon 6, n=143 | -1.8 (11.47)
  St DBP Mon 9, n=125 | -1.9 (10.17)
  St DBP Mon 12, n=170 | -1.0 (11.18)
  St DBP Mon 16, n=104 | -1.8 (11.14)
  St DBP Mon 20, n=100 | -1.0 (12.02)
  St DBP Mon 24, n=110 | 0.5 (11.78)
  St DBP Mon 28, n=87 | -1.0 (12.83)
  St DBP Mon 32, n=84 | 0.9 (11.95)
  St DBP Mon 36, n=91 | -0.7 (10.78)
  St DBP Mon 40, n=77 | -0.6 (11.09)
  St DBP Mon 44, n=75 | -0.6 (11.67)
  St DBP Mon 48, n=81 | 0.1 (11.74)
  St DBP Mon 52, n=67 | 1.0 (11.49)
  St DBP Mon 56, n=62 | -1.0 (11.2)
  St DBP Mon 60, n=69 | -1.9 (14.12)
  St DBP Mon 64, n=49 | -2.1 (11.94)
  St DBP Mon 68, n=45 | -2.9 (11.91)
  St DBP Mon 72, n=56 | 0.5 (11.13)
  St DBP Mon 76, n=30 | -2.4 (13.08)
  St DBP Mon 80, n=23 | -2.0 (10.86)
  St DBP Mon 84, n=34 | -0.6 (12.17)
  St DBP Mon 88, n=17 | 0.6 (8.99)
  St DBP Mon 92, n=16 | -3.1 (9.84)
  St DBP Mon 96, n=19 | 2.3 (8.81)
  St DBP Mon 100, n=7 | -4.9 (4.41)
  St DBP Mon 104, n=1 | -20.0 (NA) — Standard deviation value was not available as only one participant was analyzed
  St DBP Mon 108, n=10 | -4.5 (5.46)
  Su SBP Mon 1, n=173 | -1.1 (14.70)
  Su SBP Mon 3, n=159 | 0.3 (12.96)
  Su SBP Mon 6, n=143 | -0.7 (14.78)
  Su SBP Mon 9, n=125 | -0.4 (14.14)
  Su SBP Mon 12, n=173 | 0.4 (15.70)
  Su SBP Mon 16, n=104 | -2.2 (15.08)
  Su SBP Mon 20, n=100 | -0.7 (15.62)
  Su SBP Mon 24, n=112 | 0.5 (16.11)
  Su SBP Mon 28, n=88 | -0.1 (16.06)
  Su SBP Mon 32, n=85 | 0.3 (16.57)
  Su SBP Mon 36, n=92 | 0.3 (15.78)
  Su SBP Mon 40, n=78 | -0.8 (15.08)
  Su SBP Mon 44, n=76 | 0.3 (16.62)
  Su SBP Mon 48, n=82 | 2.6 (15.99)
  Su SBP Mon 52, n=68 | 3.3 (15.32)
  Su SBP Mon 56, n=63 | 1.3 (15.30)
  Su SBP Mon 60, n=70 | 0.7 (13.57)
  Su SBP Mon 64, n=50 | 0.1 (18.76)
  Su SBP Mon 68, n=45 | -0.2 (18.29)
  Su SBP Mon 72, n=57 | 0.8 (17.21)
  Su SBP Mon 76, n=31 | -1.2 (17.42)
  Su SBP Mon 80, n=24 | -2.6 (12.80)
  Su SBP Mon 84, n=36 | -3.0 (18.16)
  Su SBP Mon 88, n=17 | 0.6 (12.07)
  Su SBP Mon 92, n=16 | -0.9 (17.07)
  Su SBP Mon 96, n=19 | -0.9 (12.33)
  Su SBP Mon 100, n=7 | -3.6 (9.95)
  Su SBP Mon 104, n=1 | -20.0 (NA) — Standard deviation value was not available as only one participant was analyzed
  Su SBP Mon 108, n=10 | -4.4 (16.60)
  St SBP Mon 1, n=173 | 0.3 (14.10)
  St SBP Mon 3, n=159 | -1.6 (15.38)
  St SBP Mon 6, n=143 | 0.1 (14.35)
  St SBP Mon 9, n=125 | 0.2 (14.84)
  St SBP Mon 12, n=170 | 1.4 (15.25)
  St SBP Mon 16, n=104 | 0.1 (14.69)
  St SBP Mon 20, n=100 | 2.1 (16.05)
  St SBP Mon 24, n=110 | 3.8 (17.42)
  St SBP Mon 28, n=87 | 1.6 (15.53)
  St SBP Mon 32, n=84 | 3.1 (17.06)
  St SBP Mon 36, n=91 | 1.7 (15.20)
  St SBP Mon 40, n=77 | 1.7 (16.79)
  St SBP Mon 44, n=75 | 2.7 (15.80)
  St SBP Mon 48, n=81 | 3.3 (14.51)
  St SBP Mon 52, n=67 | 3.9 (18.37)
  St SBP Mon 56, n=62 | 2.7 (13.99)
  St SBP Mon 60, n=69 | 2.1 (13.41)
  St SBP Mon 64, n=49 | 2.4 (17.27)
  St SBP Mon 68, n=45 | -0.3 (15.98)
  St SBP Mon 72, n=56 | 2.3 (17.23)
  St SBP Mon 76, n=30 | -4.5 (17.63)
  St SBP Mon 80, n=23 | -1.1 (13.70)
  St SBP Mon 84, n=34 | -1.9 (13.46)
  St SBP Mon 88, n=17 | 2.1 (11.89)
  St SBP Mon 92, n=16 | -4.9 (14.38)
  St SBP Mon 96, n=19 | 0.5 (12.24)
  St SBP Mon 100, n=7 | -4.6 (11.16)
  St SBP Mon 104, n=1 | -22.0 (NA) — Standard deviation value was not available as only one participant was analyzed
  St SBP Mon 108, n=10 | -5.5 (7.14)

5. Primary Outcome: Change From Baseline in Heart Rate
Description: Heart rate (HR) was measured in supine (Su) position and again in standing (St) position after the participant was standing for approximately 2 minutes at each study visit (Month 1, Month 3, Month 6, Month 9, Month 12 and every 4 months after Month 12). Baseline assessment in this study is defined as the last assessment for the endpoint in parent study taken prior to the first active treatment with Retigabine. Change from Baseline was calculated as post-Baseline value minus Baseline value. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles). NA indicates that data were not available.
Time Frame: Baseline and Up to Month 108
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Beats per Minute
Arm/Group | Overall Study
Number analyzed (Participants) | 181
Beats per Minute
  Su HR Mon 1, n=174 | -1.0 (10.21)
  Su HR Mon 3, n=159 | -0.7 (11.34)
  Su HR Mon 6, n=143 | -0.2 (11.57)
  Su HR Mon 9, n=124 | -1.0 (11.33)
  Su HR Mon 12, n=173 | -0.1 (12.02)
  Su HR Mon 16, n=104 | 1.1 (12.51)
  Su HR Mon 20, n=100 | 1.1 (12.10)
  Su HR Mon 24, n=112 | -0.1 (15.92)
  Su HR Mon 28, n=88 | -0.8 (13.11)
  Su HR Mon 32, n=85 | 0.4 (12.56)
  Su HR Mon 36, n=92 | -1.7 (11.38)
  Su HR Mon 40, n=78 | -0.6 (13.28)
  Su HR Mon 44, n=76 | -2.8 (12.47)
  Su HR Mon 48, n=82 | -2.1 (11.25)
  Su HR Mon 52, n=67 | -1.5 (11.39)
  Su HR Mon 56, n=63 | -1.8 (12.30)
  Su HR Mon 60, n=70 | -1.2 (12.89)
  Su HR Mon 64, n=50 | -2.1 (11.54)
  Su HR Mon 68, n=45 | 1.2 (13.87)
  Su HR Mon 72, n=57 | -1.9 (12.32)
  Su HR Mon 76, n=31 | -1.6 (13.05)
  Su HR Mon 80, n=24 | -2.2 (11.93)
  Su HR Mon 84, n=36 | -2.4 (12.56)
  Su HR Mon 88, n=17 | 1.5 (13.98)
  Su HR Mon 92, n=16 | -2.7 (11.52)
  Su HR Mon 96, n=19 | -1.0 (14.35)
  Su HR Mon 100, n=7 | -8.3 (19.10)
  Su HR Mon 104, n=1 | -6.0 (NA) — Standard Deviation value was not available as only one participant was analyzed
  Su HR Mon 108, n=10 | -3.4 (12.86)
  St HR Mon 1, n=174 | 0.7 (11.97)
  St HR Mon 3, n=158 | 1.0 (12.02)
  St HR Mon 6, n=143 | 1.6 (12.82)
  St HR Mon 9, n=124 | 1.1 (12.99)
  St HR Mon 12, n=170 | 2.3 (12.64)
  St HR Mon 16, n=104 | 2.5 (12.71)
  St HR Mon 20, n=100 | 0.2 (13.35)
  St HR Mon 24, n=110 | 2.6 (17.38)
  St HR Mon 28, n=87 | -0.8 (13.79)
  St HR Mon 32, n=84 | 1.7 (11.71)
  St HR Mon 36, n=91 | -0.4 (12.40)
  St HR Mon 40, n=77 | 0.4 (11.51)
  St HR Mon 44, n=75 | -0.3 (12.74)
  St HR Mon 48, n=81 | -1.9 (12.57)
  St HR Mon 52, n=67 | -0.3 (12.71)
  St HR Mon 56, n=62 | 1.3 (12.21)
  St HR Mon 60, n=69 | -0.2 (14.44)
  St HR Mon 64, n=49 | 1.3 (14.29)
  St HR Mon 68, n=45 | 4.1 (14.77)
  St HR Mon 72, n=56 | 0.4 (12.10)
  St HR Mon 76, n=30 | 1.9 (13.26)
  St HR Mon 80, n=23 | 3.0 (11.81)
  St HR Mon 84, n=35 | 0.2 (13.24)
  St HR Mon 88, n=17 | 3.6 (12.24)
  St HR Mon 92, n=16 | 3.1 (10.13)
  St HR Mon 96, n=19 | 3.2 (13.12)
  St HR Mon 100, n=7 | 2.6 (10.72)
  St HR Mon 104, n=1 | 0.0 (NA) — Standard Deviation value was not available as only one participant was analyzed
  St HR Mon 108, n=10 | -5.4 (11.37)

6. Primary Outcome: Change From Baseline in Body Temperature
Description: Body temperature was measured in degree Celsius at each study visit (Month 1, Month 3, Month 6, Month 9, Month 12 and every 4 months after Month 12). Baseline assessment in this study is defined as the last assessment for the endpoint in parent study taken prior to the first active treatment with Retigabine. Change from Baseline was calculated as post-Baseline value minus Baseline value. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles). NA indicates that data were not available
Time Frame: Baseline and Up to Month 108
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | Overall Study
Number analyzed (Participants) | 181
Degree Celsius
  Temperature, Mon 1, n=174 | -0.04 (0.437)
  Temperature, Mon 3, n=158 | -0.08 (0.460)
  Temperature, Mon 6, n=142 | -0.05 (0.455)
  Temperature, Mon 9, n=124 | -0.06 (0.479)
  Temperature, Mon 12, n=172 | -0.07 (0.489)
  Temperature, Mon 16, n=102 | -0.01 (0.477)
  Temperature, Mon 20, n=98 | -0.00 (0.495)
  Temperature, Mon 24, n=110 | -0.07 (0.532)
  Temperature, Mon 28, n=86 | -0.08 (0.457)
  Temperature, Mon 32, n=85 | -0.09 (0.456)
  Temperature, Mon 36, n=92 | -0.13 (0.543)
  Temperature, Mon 40, n=77 | -0.12 (0.492)
  Temperature, Mon 44, n=76 | -0.07 (0.523)
  Temperature, Mon 48, n=82 | -0.06 (0.525)
  Temperature, Mon 52, n=68 | -0.13 (0.439)
  Temperature, Mon 56, n=63 | -0.09 (0.566)
  Temperature, Mon 60, n=70 | -0.02 (0.436)
  Temperature, Mon 64, n=48 | -0.12 (0.451)
  Temperature, Mon 68, n=45 | -0.01 (0.497)
  Temperature, Mon 72, n=57 | -0.06 (0.433)
  Temperature, Mon 76, n=31 | -0.04 (0.506)
  Temperature, Mon 80, n=24 | -0.08 (0.472)
  Temperature, Mon 84, n=36 | -0.19 (0.481)
  Temperature, Mon 88, n=17 | -0.20 (0.496)
  Temperature, Mon 92, n=16 | -0.14 (0.542)
  Temperature, Mon 96, n=19 | -0.26 (0.512)
  Temperature, Mon 100, n=7 | -0.14 (0.690)
  Temperature, Mon 104, n=1 | 1.00 (NA) — Standard Deviation value was not available as only one participant was analyzed
  Temperature, Mon 108, n=10 | -0.15 (0.645)

7. Primary Outcome: Change From Baseline in Weight
Description: Weight was measured in ordinary indoor clothing (without shoes) and was recorded at each study visit (On Month 1, Month 3, Month 6, Month 9, Month 12 and every 4 months after Month 12). Baseline assessment in this study is defined as the last assessment for the endpoint in parent study taken prior to the first active treatment with Retigabine. Change from Baseline was calculated as post-Baseline value minus Baseline value. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles). NA indicates that data were not available.
Time Frame: Baseline and Up to Month 108
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Kilograms
Groups:
- Overall Study: Participants received retigabine tablets for a total dose of between 600 to 1200 mg/day (dose administered twice daily or TID) an adjunct therapy to their ongoing antiepileptic drugs with or without vagal nerve stimulation treatment until withdrawal, withdrawn consent or switched to commercial product.
Arm/Group | Overall Study
Number analyzed (Participants) | 181
Kilograms
  Weight, Mon 1, n=172 | 1.94 (3.691)
  Weight, Mon 3, n=159 | 1.85 (6.455)
  Weight, Mon 6, n=143 | 1.68 (5.315)
  Weight, Mon 9, n=123 | 1.57 (6.149)
  Weight, Mon 12, n=171 | 1.31 (6.961)
  Weight, Mon 16, n=104 | 2.17 (8.799)
  Weight, Mon 20, n=101 | 1.62 (7.786)
  Weight, Mon 24, n=111 | 1.21 (8.178)
  Weight, Mon 28, n=88 | 0.35 (8.859)
  Weight, Mon 32, n=85 | 0.07 (9.084)
  Weight, Mon 36, n=92 | 0.61 (8.066)
  Weight, Mon 40, n=78 | 0.84 (9.106)
  Weight, Mon 44, n=76 | 0.88 (8.137)
  Weight, Mon 48, n=82 | 0.73 (9.097)
  Weight, Mon 52, n=68 | 1.10 (9.401)
  Weight, Mon 56, n=62 | 1.28 (8.998)
  Weight, Mon 60, n=69 | 0.94 (9.335)
  Weight, Mon 64, n=49 | 2.13 (10.004)
  Weight, Mon 68, n=44 | 2.77 (9.79)
  Weight, Mon 72, n=57 | 0.85 (10.701)
  Weight, Mon 76, n=31 | 3.30 (8.260)
  Weight, Mon 80, n=24 | 1.48 (7.899)
  Weight, Mon 84, n=36 | 2.47 (10.022)
  Weight, Mon 88, n=17 | 1.45 (9.036)
  Weight, Mon 92, n=16 | 1.64 (7.571)
  Weight, Mon 96, n=19 | 0.48 (9.380)
  Weight, Mon 100, n=7 | 4.31 (7.006)
  Weight, Mon 104, n=1 | 2.10 (NA) — Standard Deviation value was not available as only one participant was analyzed
  Weight, Mon 108, n=10 | 3.18 (5.743)

8. Primary Outcome: Change From Baseline in the 12-lead Electrocardiogram (ECG) Parameters-PR Interval, QRS Duration, Uncorrected QT (uQT) Interval, Corrected QT (Bazett's Correction) Interval (QTcB), Corrected QT (Friedericia's Correction) Interval (QTcF)
Description: A 12-lead ECG was performed at each study visit during the first year of the study (Month 1, Month 3, Month 6, Month 9, Month 12) and annually after one year. The following electrocardiogram parameters are presented PR Interval, QRS Duration, Uncorrected QT interval (uQT), Corrected QT (Bazett's correction) interval (QTcB), Corrected QT (Friedericia's correction) interval (QTcF). Baseline assessment in this study is defined as the last assessment for the endpoint in parent study taken prior to the first active treatment with Retigabine. Change from Baseline was calculated as post-Baseline value minus Baseline value. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles). NA indicates that data were not available.
Time Frame: Baseline and Up to Month 108
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Milliseconds (msec)
Groups:
- Overall Study Arm: Participants received retigabine tablets for a total dose of between 600 to 1200 mg/day (dose administered twice daily or TID) an adjunct therapy to their ongoing antiepileptic drugs with or without vagal nerve stimulation treatment until withdrawal, withdrawn consent or switched to commercial product.
Arm/Group | Overall Study Arm
Number analyzed (Participants) | 181
Milliseconds (msec)
  QTcB, Mon 1, n=172 | 3.3 (18.13)
  QTcB, Mon 3, n=157 | 5.8 (18.84)
  QTcB, Mon 6, n=139 | 1.5 (17.29)
  QTcB, Mon 9, n=121 | 2.2 (17.18)
  QTcB, Mon 12, n=168 | 5.7 (19.18)
  QTcB, Mon 24, n=109 | 5.9 (18.52)
  QTcB, Mon 36, n=89 | 3.7 (20.32)
  QTcB, Mon 48, n=80 | 5.4 (17.74)
  QTcB, Mon 60, n=70 | 5.1 (17.76)
  QTcB, Mon 72, n=54 | 5.5 (15.86)
  QTcB, Mon 84, n=36 | 8.1 (16.02)
  QTcB, Mon 96, n=19 | 11.0 (15.95)
  QTcB, Mon 108, n=10 | -3.7 (17.25)
  QTcF, Mon 1, n=172 | 4.7 (16.12)
  QTcF, Mon 3, n=157 | 6.0 (16.57)
  QTcF, Mon 6, n=139 | 1.4 (15.79)
  QTcF, Mon 9, n=121 | 2.9 (15.57)
  QTcF, Mon 12, n=168 | 5.5 (16.51)
  QTcF, Mon 24, n=109 | 4.7 (15.91)
  QTcF, Mon 36, n=89 | 4.3 (16.58)
  QTcF, Mon 48, n=80 | 5.9 (14.93)
  QTcF, Mon 60, n=70 | 5.9 (13.94)
  QTcF, Mon 72, n=54 | 7.2 (16.89)
  QTcF, Mon 84, n=36 | 9.3 (14.20)
  QTcF, Mon 96, n=19 | 8.9 (14.83)
  QTcF, Mon 108, n=10 | -5.7 (12.64)
  PR interval, Mon 1, n=173 | -0.8 (13.07)
  PR interval, Mon 3, n=158 | 1.0 (12.99)
  PR interval, Mon 6, n=139 | 0.0 (12.69)
  PR interval, Mon 9, n=123 | -1.4 (12.44)
  PR interval, Mon 12, n=168 | -1.0 (12.61)
  PR interval, Mon 24, n=110 | -3.1 (12.16)
  PR interval, Mon 36, n=89 | -0.3 (11.39)
  PR interval, Mon 48, n=80 | 0.3 (16.32)
  PR interval, Mon 60, n=71 | 2.5 (14.12)
  PR interval, Mon 72, n=53 | 2.2 (11.71)
  PR interval, Mon 84, n=36 | 4.3 (9.34)
  PR interval, Mon 96, n=19 | -2.4 (13)
  PR interval, Mon 108, n=10 | 0.0 (15.5)
  QRS duration, Mon 1, n=174 | 0.4 (7.37)
  QRS duration, Mon 3, n=159 | -0.2 (7.64)
  QRS duration, Mon 6, n=142 | -0.2 (7.05)
  QRS duration, Mon 9, n=124 | 0.4 (8.04)
  QRS duration, Mon 12, n=171 | -0.0 (9.4)
  QRS duration, Mon 24, n=112 | 0.7 (8.56)
  QRS duration, Mon 36, n=90 | 1.6 (7.31)
  QRS duration, Mon 48, n=81 | 4.0 (7.82)
  QRS duration, Mon 60, n=70 | 3.9 (8.19)
  QRS duration, Mon 72, n=55 | 6.2 (9.15)
  QRS duration, Mon 84, n=36 | 4.2 (7.94)
  QRS duration, Mon 96, n=19 | 3.8 (7.21)
  QRS duration, Mon 108, n=10 | 3.7 (9.4)
  uQT, Mon 1, n=172 | 7.5 (22.93)
  uQT, Mon 3, n=157 | 6.4 (25.31)
  uQT, Mon 6, n=139 | 1.4 (25.95)
  uQT, Mon 9, n=121 | 4.3 (25.00)
  uQT, Mon 12, n=168 | 5.1 (24.70)
  uQT, Mon 24, n=109 | 2.8 (23.97)
  uQT, Mon 36, n=89 | 5.5 (22.57)
  uQT, Mon 48, n=80 | 7.2 (22.42)
  uQT, Mon 60, n=70 | 7.3 (24.74)
  uQT, Mon 72, n=54 | 11.0 (28.33)
  uQT, Mon 84, n=36 | 12.5 (26.56)
  uQT, Mon 96, n=19 | 5.4 (26.73)
  uQT, Mon 108, n=10 | -8.7 (14.01)

9. Primary Outcome: Change From Baseline in the 12-lead Electrocardiogram (ECG) Parameter-RR Interval
Description: A 12-lead ECG was performed at each study visit during the first year of the study (Month 1, Month 3, Month 6, Month 9, Month 12) and annually after one year. The following electrocardiogram parameters are presented: RR Interval. Baseline assessment in this study is defined as the last assessment for the endpoint in parent study taken prior to the first active treatment with Retigabine. Change from Baseline was calculated as post-Baseline value minus Baseline value. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline and Up to Month 108
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Seconds (sec)
Arm/Group | Overall Study Arm
Number analyzed (Participants) | 181
Seconds (sec)
  RR interval, Mon 1, n=174 | 0.0195 (0.11576)
  RR interval, Mon 3, n=159 | 0.0029 (0.12883)
  RR interval, Mon 6, n=142 | -0.0007 (0.13151)
  RR interval, Mon 9, n=124 | 0.0103 (0.12659)
  RR interval, Mon 12, n=172 | -0.0015 (0.12556)
  RR interval, Mon 24, n=112 | -0.0119 (0.1206)
  RR interval, Mon 36, n=92 | 0.0144 (0.12476)
  RR interval, Mon 48, n=81 | 0.0145 (0.12175)
  RR interval, Mon 60, n=71 | 0.0098 (0.14452)
  RR interval, Mon 72, n=55 | 0.0251 (0.12713)
  RR interval, Mon 84, n=36 | 0.0285 (0.15006)
  RR interval, Mon 96, n=19 | -0.0237 (0.1485)
  RR interval, Mon 108, n=10 | -0.0173 (0.10885)

10. Primary Outcome: Change From Baseline in Electrocardiogram (ECG) Parameter-QRS Axis
Description: A 12-lead ECG was performed at each study visit during the first year of the study (Month 1, Month 3, Month 6, Month 9, Month 12) and annually after one year. ECG parameter QRS Axis is presented here. Baseline assessment in this study is defined as the last assessment for the endpoint in parent study taken prior to the first active treatment with Retigabine. Change from Baseline was calculated as post-Baseline value minus Baseline value. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline and Up to Month 108
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Degree
Groups:
- Overall Study Arm: Participants received retigabine tablets for a total dose of between 600 to 1200 mg/day (dose administered twice daily or TID) as an adjunct therapy to their ongoing antiepileptic drugs with or without vagal nerve stimulation treatment until withdrawal, withdrawn consent or switched to commercial product.
Arm/Group | Overall Study Arm
Number analyzed (Participants) | 181
Degree
  QRS axis, Mon 1, n=167 | -1.3 (14.34)
  QRS axis, Mon 3, n=151 | -2.9 (15.94)
  QRS axis, Mon 6, n=134 | -1.5 (11.50)
  QRS axis, Mon 9, n=118 | -2.3 (11.8)
  QRS axis, Mon 12, n=160 | -3.1 (13.72)
  QRS axis, Mon 24, n=104 | -1.9 (13.03)
  QRS axis, Mon 36, n=87 | -2.5 (11.43)
  QRS axis, Mon 48, n=77 | -3.4 (19.82)
  QRS axis, Mon 60, n=68 | -8.0 (14.50)
  QRS axis, Mon 72, n=52 | -4.0 (12.31)
  QRS axis, Mon 84, n=34 | -4.1 (16.09)
  QRS axis, Mon 96, n=18 | -4.9 (8.53)
  QRS axis, Mon 108, n=10 | -7.0 (8.81)

11. Primary Outcome: Change From Baseline in Hematology Parameters- Bands, Basophils, Eosinophils, Lymphocytes, Metamyelocyte, Monocytes, Neutrophils, Platelets, White Blood Cells Count (WBC)
Description: Following hematology parameters were assessed, Bands (Band neutrophils), Basophils, Eosinophils, Lymphocytes, Metamyelocyte, Monocytes, Neutrophils, Platelets and WBC. Hematology parameters were assessed at Month 1, Month 2, Month 3, Month 6, Month 8, Month 9, Month 10, Month 12 and every 4 months after Month 12. Baseline assessment in this study is defined as the last assessment for the endpoint in parent study taken prior to the first active treatment with Retigabine. Change from Baseline was calculated as post-Baseline value minus Baseline value. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles). NA indicates that data were not available.
Time Frame: Baseline and Up to Month 108
Population: Safety Population
Measure: Mean (Standard Deviation); unit: 10^9 cells/Liter
Arm/Group | Overall Study Arm
Number analyzed (Participants) | 181
10^9 cells/Liter
  Bands, Mon 1, n=2 | -0.135 (0.1768)
  Bands, Mon 9, n=2 | -0.205 (0.6576)
  Bands, Mon 20, n=2 | -0.095 (0.1202)
  Basophils, Mon 1, n=168 | -0.001 (0.0270)
  Basophils, Mon 2, n=15 | -0.015 (0.0307)
  Basophils, Mon 3, n=153 | 0.001 (0.0274)
  Basophils, Mon 4, n=26 | -0.002 (0.0199)
  Basophils, Mon 6, n=137 | 0.004 (0.0245)
  Basophils, Mon 8, n=42 | 0.002 (0.0258)
  Basophils, Mon 9, n=121 | 0.003 (0.0274)
  Basophils, Mon 10, n=54 | 0.001 (0.0241)
  Basophils, Mon 12, n=165 | 0.001 (0.0298)
  Basophils, Mon 16, n=96 | 0.005 (0.0288)
  Basophils, Mon 20, n=92 | 0.004 (0.0271)
  Basophils, Mon 24, n=109 | 0.008 (0.0289)
  Basophils, Mon 28, n=84 | 0.005 (0.0289)
  Basophils, Mon 32, n=81 | 0.005 (0.0301)
  Basophils, Mon 36, n=91 | 0.006 (0.0295)
  Basophils, Mon 40, n=74 | 0.004 (0.0243)
  Basophils, Mon 44, n=72 | 0.004 (0.0200)
  Basophils, Mon 48, n=77 | 0.004 (0.0313)
  Basophils, Mon 52, n=65 | -0.004 (0.0227)
  Basophils, Mon 56, n=63 | -0.004 (0.0234)
  Basophils, Mon 60, n=71 | -0.003 (0.0238)
  Basophils, Mon 64, n=49 | -0.003 (0.0195)
  Basophils, Mon 68, n=43 | 0.001 (0.0197)
  Basophils, Mon 72, n=53 | -0.003 (0.0227)
  Basophils, Mon 76, n=31 | -0.000 (0.0218)
  Basophils, Mon 80, n=24 | -0.001 (0.0198)
  Basophils, Mon 84, n=33 | 0.002 (0.0238)
  Basophils, Mon 88, n=16 | 0.003 (0.0202)
  Basophils, Mon 92, n=15 | 0.005 (0.0288)
  Basophils, Mon 96, n=19 | 0.006 (0.0257)
  Basophils, Mon 100, n=7 | 0.021 (0.0157)
  Basophils, Mon 104, n=1 | -0.020 (NA) — Standard deviation value was not available as only one participant was analyzed
  Basophils, Mon 108, n=10 | 0.012 (0.0210)
  Eosinophils, Mon 1, n=168 | -0.008 (0.1009)
  Eosinophils, Mon 2, n=15 | 0.023 (0.0948)
  Eosinophils, Mon 3, n=153 | -0.010 (0.1329)
  Eosinophils, Mon 4, n=26 | -0.003 (0.1236)
  Eosinophils, Mon 6, n=137 | -0.015 (0.1208)
  Eosinophils, Mon 8, n=42 | -0.022 (0.1078)
  Eosinophils, Mon 9, n=121 | -0.010 (0.1166)
  Eosinophils, Mon 10, n=54 | 0.000 (0.1083)
  Eosinophils, Mon 12, n=165 | -0.019 (0.0943)
  Eosinophils, Mon 16, n=96 | -0.006 (0.1145)
  Eosinophils, Mon 20, n=92 | -0.009 (0.0941)
  Eosinophils, Mon 24, n=109 | -0.002 (0.1108)
  Eosinophils, Mon 28, n=84 | -0.016 (0.1114)
  Eosinophils, Mon 32, n=81 | 0.001 (0.1192)
  Eosinophils, Mon 36, n=91 | -0.006 (0.1026)
  Eosinophils, Mon 40, n=74 | -0.004 (0.1165)
  Eosinophils, Mon 44, n=72 | -0.014 (0.1158)
  Eosinophils, Mon 48, n=77 | -0.002 (0.1230)
  Eosinophils, Mon 52, n=65 | -0.011 (0.1137)
  Eosinophils, Mon 56, n=63 | -0.002 (0.1251)
  Eosinophils, Mon 60, n=71 | -0.014 (0.1123)
  Eosinophils, Mon 64, n=49 | -0.008 (0.0989)
  Eosinophils, Mon 68, n=43 | -0.000 (0.1122)
  Eosinophils, Mon 72, n=53 | 0.005 (0.1049)
  Eosinophils, Mon 76, n=31 | -0.003 (0.1102)
  Eosinophils, Mon 80, n=24 | -0.010 (0.0837)
  Eosinophils, Mon 84, n=33 | -0.000 (0.1105)
  Eosinophils, Mon 88, n=16 | 0.030 (0.0602)
  Eosinophils, Mon 92, n=15 | 0.006 (0.0631)
  Eosinophils, Mon 96, n=19 | 0.018 (0.0511)
  Eosinophils, Mon 100, n=7 | 0.033 (0.093)
  Eosinophils, Mon 104, n=1 | 0.030 (NA) — Standard deviation value was not available as only one participant was analyzed
  Eosinophils, Mon 108, n=10 | -0.005 (0.0792)
  Lymphocytes, Mon 1, n=168 | -0.178 (0.4512)
  Lymphocytes, Mon 2, n=15 | -0.043 (0.6364)
  Lymphocytes, Mon 3, n=153 | -0.134 (0.4336)
  Lymphocytes, Mon 4, n=26 | 0.054 (0.3529)
  Lymphocytes, Mon 6, n=137 | -0.055 (0.4415)
  Lymphocytes, Mon 8, n=42 | 0.168 (0.7157)
  Lymphocytes, Mon 9, n=121 | -0.031 (0.472)
  Lymphocytes, Mon 10, n=54 | 0.120 (0.5265)
  Lymphocytes, Mon 12, n=165 | 0.009 (0.5438)
  Lymphocytes, Mon 16, n=96 | -0.053 (0.5393)
  Lymphocytes, Mon 20, n=92 | -0.031 (0.5364)
  Lymphocytes, Mon 24, n=109 | -0.069 (0.4973)
  Lymphocytes, Mon 28, n=84 | -0.077 (0.5271)
  Lymphocytes, Mon 32, n=81 | 0.013 (0.5920)
  Lymphocytes, Mon 36, n=91 | -0.055 (0.4798)
  Lymphocytes, Mon 40, n=74 | -0.028 (0.4699)
  Lymphocytes, Mon 44, n=72 | 0.008 (0.4681)
  Lymphocytes, Mon 48, n=77 | 0.061 (0.5921)
  Lymphocytes, Mon 52, n=65 | -0.049 (0.4875)
  Lymphocytes, Mon 56, n=63 | -0.065 (0.5298)
  Lymphocytes, Mon 60, n=71 | -0.025 (0.5503)
  Lymphocytes, Mon 64, n=49 | -0.011 (0.5106)
  Lymphocytes, Mon 68, n=43 | -0.002 (0.6027)
  Lymphocytes, Mon 72, n=53 | -0.052 (0.5410)
  Lymphocytes, Mon 76, n=31 | 0.104 (0.6589)
  Lymphocytes, Mon 80, n=24 | 0.149 (0.6626)
  Lymphocytes, Mon 84, n=33 | 0.154 (0.6009)
  Lymphocytes, Mon 88, n=16 | 0.189 (0.4887)
  Lymphocytes, Mon 92, n=15 | 0.405 (0.5963)
  Lymphocytes, Mon 96, n=19 | 0.285 (0.6170)
  Lymphocytes, Mon 100, n=7 | 0.144 (0.4465)
  Lymphocytes, Mon 104, n=1 | 0.000 (NA) — Standard deviation value was not available as only one participant was analyzed
  Lymphocytes, Mon 108, n=10 | 0.044 (0.5883)
  Metamyelocyte, Mon 3, n=1 | -0.010 (NA) — Standard deviation value was not available as only one participant was analyzed
  Monocytes, Mon 1, n=168 | 0.006 (0.1755)
  Monocytes, Mon 2, n=15 | 0.002 (0.2583)
  Monocytes, Mon 3, n=153 | 0.016 (0.1730)
  Monocytes, Mon 4, n=26 | 0.039 (0.1759)
  Monocytes, Mon 6, n=137 | -0.001 (0.1628)
  Monocytes, Mon 8, n=42 | 0.033 (0.2000)
  Monocytes, Mon 9, n=121 | -0.002 (0.1808)
  Monocytes, Mon 10, n=54 | 0.029 (0.1686)
  Monocytes, Mon 12, n=165 | -0.007 (0.1724)
  Monocytes, Mon 16, n=96 | -0.021 (0.1651)
  Monocytes, Mon 20, n=92 | -0.009 (0.1573)
  Monocytes, Mon 24, n=109 | -0.004 (0.2189)
  Monocytes, Mon 28, n=84 | -0.031 (0.1759)
  Monocytes, Mon 32, n=81 | -0.005 (0.1673)
  Monocytes, Mon 36, n=91 | -0.039 (0.1821)
  Monocytes, Mon 40, n=74 | -0.013 (0.1718)
  Monocytes, Mon 44, n=72 | -0.037 (0.1807)
  Monocytes, Mon 48, n=77 | -0.036 (0.1869)
  Monocytes, Mon 52, n=65 | -0.026 (0.1743)
  Monocytes, Mon 56, n=63 | -0.035 (0.1776)
  Monocytes, Mon 60, n=71 | -0.013 (0.1720)
  Monocytes, Mon 64, n=49 | -0.024 (0.1486)
  Monocytes, Mon 68, n=43 | 0.003 (0.1491)
  Monocytes, Mon 72, n=53 | -0.007 (0.1704)
  Monocytes, Mon 76, n=31 | 0.038 (0.1456)
  Monocytes, Mon 80, n=24 | 0.019 (0.1473)
  Monocytes, Mon 84, n=33 | 0.065 (0.1555)
  Monocytes, Mon 88, n=16 | -0.006 (0.1699)
  Monocytes, Mon 92, n=15 | 0.029 (0.1737)
  Monocytes, Mon 96, n=19 | 0.035 (0.1437)
  Monocytes, Mon 100, n=7 | 0.004 (0.1274)
  Monocytes, Mon 104, n=1 | 0.070 (NA) — Standard deviation value was not available as only one participant was analyzed
  Monocytes, Mon 108, n=10 | 0.064 (0.2400)
  Neutrophils, Mon 1, n=168 | 0.158 (1.5462)
  Neutrophils, Mon 2, n=15 | -0.500 (1.6917)
  Neutrophils, Mon 3, n=153 | 0.211 (1.2173)
  Neutrophils, Mon 4, n=26 | -0.003 (1.1181)
  Neutrophils, Mon 6, n=137 | 0.124 (1.0916)
  Neutrophils, Mon 8, n=42 | -0.427 (1.1287)
  Neutrophils, Mon 9, n=121 | 0.074 (1.0966)
  Neutrophils, Mon 10, n=54 | 0.211 (1.4455)
  Neutrophils, Mon 12, n=165 | 0.309 (1.2657)
  Neutrophils, Mon 16, n=96 | 0.232 (1.0227)
  Neutrophils, Mon 20, n=92 | 0.145 (1.039)
  Neutrophils, Mon 24, n=109 | 0.221 (1.1556)
  Neutrophils, Mon 28, n=84 | -0.032 (1.1173)
  Neutrophils, Mon 32, n=81 | -0.034 (1.1604)
  Neutrophils, Mon 36, n=91 | -0.054 (1.0499)
  Neutrophils, Mon 40, n=74 | 0.141 (1.101)
  Neutrophils, Mon 44, n=72 | 0.003 (1.0641)
  Neutrophils, Mon 48, n=77 | 0.197 (1.4174)
  Neutrophils, Mon 56, n=63 | 0.075 (1.069)
  Neutrophils, Mon 52, n=65 | 0.151 (1.1449)
  Neutrophils, Mon 60, n=71 | 0.203 (1.653)
  Neutrophils, Mon 64, n=49 | -0.042 (1.0603)
  Neutrophils, Mon 68, n=43 | 0.304 (1.3417)
  Neutrophils, Mon 72, n=53 | 0.337 (1.3877)
  Neutrophils, Mon 76, n=31 | 0.380 (0.9556)
  Neutrophils, Mon 80, n=24 | 0.495 (1.1337)
  Neutrophils, Mon 84, n=33 | 0.735 (1.2746)
  Neutrophils, Mon 88, n=16 | 0.036 (0.689)
  Neutrophils, Mon 92, n=15 | 0.275 (1.2747)
  Neutrophils, Mon 96, n=19 | 0.444 (1.1230)
  Neutrophils, Mon 100, n=7 | 0.156 (0.5022)
  Neutrophils, Mon 104, n=1 | 0.270 (NA) — Standard deviation value was not available as only one participant was analyzed
  Neutrophils, Mon 108, n=10 | 0.185 (0.9415)
  Platelet Count, Mon 1, n=165 | -4.1 (38.59)
  Platelet Count, Mon 2, n=15 | 5.3 (47.49)
  Platelet Count, Mon 3, n=150 | -5.4 (40.70)
  Platelet Count, Mon 4, n=26 | -2 (54.42)
  Platelet Count, Mon 6, n=131 | -7 (48.59)
  Platelet Count, Mon 8, n=42 | 6 (49.17)
  Platelet Count, Mon 9, n=119 | -4.7 (38.65)
  Platelet Count, Mon 10, n=54 | 2.9 (39.60)
  Platelet Count, Mon 12, n=161 | -5.2 (40.72)
  Platelet Count, Mon 16, n=94 | -0.2 (46.65)
  Platelet Count, Mon 20, n=91 | -1.9 (44.44)
  Platelet Count, Mon 24, n=104 | -11.0 (42.31)
  Platelet Count, Mon 28, n=82 | -14.4 (46.60)
  Platelet Count, Mon 32, n=82 | -23.2 (45.64)
  Platelet Count, Mon 36, n=87 | -24.4 (39.19)
  Platelet Count, Mon 40, n=76 | -18.0 (40.84)
  Platelet Count, Mon 48, n=77 | -16.1 (41.68)
  Platelet Count, Mon 52, n=65 | -17.5 (35.27)
  Platelet Count, Mon 56, n=62 | -21.3 (36.88)
  Platelet Count, Mon 60, n=68 | -22.3 (38.07)
  Platelet Count, Mon 64, n=47 | -20.2 (47.45)
  Platelet Count, Mon 68, n=44 | -21.0 (48.34)
  Platelet Count, Mon 72, n=52 | -15.7 (43.17)
  Platelet Count, Mon 76, n=31 | -11.5 (52.19)
  Platelet Count, Mon 80, n=24 | -6.3 (43.84)
  Platelet Count, Mon 84, n=35 | -4.3 (40.03)
  Platelet Count, Mon 88, n=16 | -10.2 (30.96)
  Platelet Count, Mon 92, n=15 | -2.9 (25.92)
  Platelet Count, Mon 96, n=19 | -7.2 (37.84)
  Platelet Count, Mon 100, n=7 | -14.3 (50.43)
  Platelet Count, Mon 104, n=1 | -46.0 (NA) — Standard deviation value was not available as only one participant was analyzed
  Platelet Count, Mon 108, n=10 | -22.3 (40.89)
  WBC, Mon 1, n=169 | -0.00 (1.708)
  WBC, Mon 2, n=15 | -0.53 (2.281)
  WBC, Mon 3, n=154 | 0.10 (1.434)
  WBC, Mon 4, n=26 | 0.17 (1.279)
  WBC, Mon 6, n=137 | 0.06 (1.235)
  WBC, Mon 8, n=43 | -0.11 (1.577)
  WBC, Mon 9, n=122 | 0.05 (1.356)
  WBC, Mon 10, n=55 | 0.33 (1.654)
  WBC, Mon 12, n=167 | 0.30 (1.500)
  WBC, Mon 16, n=99 | 0.20 (1.362)
  WBC, Mon 20, n=96 | 0.14 (1.274)
  WBC, Mon 24, n=110 | 0.16 (1.398)
  WBC, Mon 28, n=85 | -0.14 (1.303)
  WBC, Mon 32, n=86 | 0.02 (1.347)
  WBC, Mon 36, n=91 | -0.14 (1.233)
  WBC, Mon 40, n=78 | 0.13 (1.331)
  WBC, Mon 44, n=74 | -0.04 (1.372)
  WBC, Mon 48, n=79 | 0.24 (1.438)
  WBC, Mon 52, n=68 | 0.09 (1.397)
  WBC, Mon 56, n=63 | -0.04 (1.198)
  WBC, Mon 60, n=71 | 0.18 (1.892)
  WBC, Mon 64, n=49 | -0.09 (1.236)
  WBC, Mon 68, n=44 | 0.27 (1.463)
  WBC, Mon 72, n=53 | 0.27 (1.502)
  WBC, Mon 76, n=31 | 0.51 (1.252)
  WBC, Mon 80, n=24 | 0.65 (1.219)
  WBC, Mon 84, n=35 | 0.93 (1.290)
  WBC, Mon 88, n=16 | 0.25 (0.836)
  WBC, Mon 92, n=15 | 0.73 (1.348)
  WBC, Mon 96, n=19 | 0.79 (1.129)
  WBC, Mon 100, n=7 | 0.36 (0.483)
  WBC, Mon 104, n=1 | 0.30 (NA) — Standard deviation value was not available as only one participant was analyzed
  WBC, Mon 108, n=10 | 0.31 (0.743)

12. Primary Outcome: Change From Baseline in Hematology Parameter-Red Blood Cell Count
Description: Red Blood Cell count (RBC) was assessed at Month 1, Month 2, Month 3, Month 6, Month 8, Month 9, Month 10, Month 12 and every 4 months after Month 12. Baseline assessment in this study is defined as the last assessment for the endpoint in parent study taken prior to the first active treatment with Retigabine. Change from Baseline was calculated as post-Baseline value minus Baseline value. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles). NA indicates that data were not available..
Time Frame: Baseline and Up to Month 108
Population: Safety Population
Measure: Mean (Standard Deviation); unit: 10^12 cells/Liter(L)
Arm/Group | Overall Study Arm
Number analyzed (Participants) | 181
10^12 cells/Liter(L)
  RBC, Mon 1, n=169 | -0.09 (0.281)
  RBC, Mon 2, n=15 | 0.01 (0.222)
  RBC, Mon 3, n=154 | -0.06 (0.309)
  RBC, Mon 4, n=26 | -0.16 (0.305)
  RBC, Mon 6, n=137 | -0.04 (0.287)
  RBC, Mon 8, n=43 | -0.03 (0.312)
  RBC, Mon 9, n=122 | -0.06 (0.294)
  RBC, Mon 10, n=55 | -0.01 (0.299)
  RBC, Mon 12, n=167 | 0.00 (0.291)
  RBC, Mon 16, n=99 | -0.04 (0.320)
  RBC, Mon 20, n=96 | 0.01 (0.329)
  RBC, Mon 24, n=110 | -0.01 (0.290)
  RBC, Mon 28, n=85 | -0.04 (0.324)
  RBC, Mon 32, n=86 | -0.03 (0.322)
  RBC, Mon 36, n=91 | -0.11 (0.288)
  RBC, Mon 40, n=78 | -0.11 (0.320)
  RBC, Mon 44, n=74 | -0.09 (0.318)
  RBC, Mon 48, n=79 | -0.16 (0.316)
  RBC, Mon 52, n=68 | -0.08 (0.336)
  RBC, Mon 56, n=63 | -0.13 (0.272)
  RBC, Mon 60, n=71 | -0.14 (0.317)
  RBC, Mon 64, n=49 | -0.10 (0.323)
  RBC, Mon 68, n=44 | -0.06 (0.326)
  RBC, Mon 72, n=53 | -0.09 (0.363)
  RBC, Mon 76, n=31 | 0.00 (0.373)
  RBC, Mon 80, n=24 | -0.03 (0.343)
  RBC, Mon 84, n=35 | -0.00 (0.379)
  RBC, Mon 88, n=16 | 0.03 (0.353)
  RBC, Mon 92, n=15 | 0.14 (0.300)
  RBC, Mon 96, n=19 | 0.04 (0.248)
  RBC, Mon 100, n=7 | 0.23 (0.287)
  RBC, Mon 104, n=1 | 0.30 (NA) — Standard deviation value was not available as only one participant was analyzed
  RBC, Mon 108, n=10 | 0.15 (0.207)

13. Primary Outcome: Change From Baseline in Haematocrit
Description: Haematocrit was assessed at Month 1, Month 2, Month 3, Month 6, Month 8, Month 9, Month 10, Month 12 and every 4 months after Month 12. Baseline assessment in this study is defined as the last assessment for the endpoint in parent study taken prior to the first active treatment with Retigabine. Change from Baseline was calculated as post-Baseline value minus Baseline value. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline and Up to Month 108
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Volume/Volume (v/v)
Arm/Group | Overall Study Arm
Number analyzed (Participants) | 181
Volume/Volume (v/v)
  Haematocrit, Mon 1, n=165 | -0.009 (0.0272)
  Haematocrit, Mon 2, n=15 | -0.001 (0.0210)
  Haematocrit, Mon 3, n=153 | -0.007 (0.0287)
  Haematocrit, Mon 4, n=26 | -0.012 (0.0293)
  Haematocrit, Mon 6, n=136 | -0.004 (0.0262)
  Haematocrit, Mon 8, n=41 | -0.005 (0.0248)
  Haematocrit, Mon 9, n=120 | -0.006 (0.0272)
  Haematocrit, Mon 10, n=55 | -0.002 (0.0295)
  Haematocrit, Mon 12, n=162 | -0.001 (0.0291)
  Haematocrit, Mon 16, n=98 | -0.005 (0.0292)
  Haematocrit, Mon 20, n=94 | -0.001 (0.0280)
  Haematocrit, Mon 24, n=109 | -0.002 (0.0267)
  Haematocrit, Mon 28, n=84 | -0.004 (0.0250)
  Haematocrit, Mon 32, n=85 | -0.001 (0.0273)
  Haematocrit, Mon 36, n=91 | -0.005 (0.0298)
  Haematocrit, Mon 40, n=77 | -0.004 (0.0319)
  Haematocrit, Mon 44, n=73 | -0.002 (0.0287)
  Haematocrit, Mon 48, n=76 | -0.009 (0.0376)
  Haematocrit, Mon 52, n=67 | 0.001 (0.0347)
  Haematocrit, Mon 56, n=62 | -0.001 (0.0335)
  Haematocrit, Mon 60, n=71 | 0.005 (0.0352)
  Haematocrit, Mon 64, n=49 | 0.004 (0.0332)
  Haematocrit, Mon 68, n=44 | 0.011 (0.0345)
  Haematocrit, Mon 72, n=53 | 0.008 (0.0346)
  Haematocrit, Mon 76, n=31 | 0.014 (0.0350)
  Haematocrit, Mon 80, n=23 | 0.009 (0.0272)
  Haematocrit, Mon 84, n=34 | 0.007 (0.0379)
  Haematocrit, Mon 88, n=16 | 0.017 (0.0332)
  Haematocrit, Mon 92, n=14 | 0.027 (0.0267)
  Haematocrit, Mon 96, n=18 | 0.017 (0.0311)
  Haematocrit, Mon 100, n=6 | 0.028 (0.0232)
  Haematocrit, Mon 108, n=9 | 0.030 (0.0283)

14. Primary Outcome: Change From Baseline in Haemoglobin
Description: Haemoglobin was assessed at Month 1, Month 2, Month 3, , Month 6, Month 8, Month 9, Month 10, Month 12 and every 4 months after Month 12. Baseline assessment in this study is defined as the last assessment for the endpoint in parent study taken prior to the first active treatment with Retigabine. Change from Baseline was calculated as post-Baseline value minus Baseline value. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles). NA indicates that data were not available..
Time Frame: Baseline and Up to Month 108
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Grams/Liter (g/L)
Arm/Group | Overall Study Arm
Number analyzed (Participants) | 181
Grams/Liter (g/L)
  Haemoglobin, Mon 1, n=169 | -3.2 (8.97)
  Haemoglobin, Mon 2, n=15 | -0.9 (7.26)
  Haemoglobin, Mon 3, n=154 | -2.6 (9.41)
  Haemoglobin, Mon 4, n=26 | -5.7 (10.44)
  Haemoglobin, Mon 6, n=137 | -2.2 (9.31)
  Haemoglobin, Mon 8, n=43 | -1.9 (9.40)
  Haemoglobin, Mon 9, n=122 | -2.9 (9.45)
  Haemoglobin, Mon 10, n=55 | -0.9 (9.26)
  Haemoglobin, Mon 12, n=167 | -0.7 (9.61)
  Haemoglobin, Mon 16, n=98 | -2.5 (9.96)
  Haemoglobin, Mon 20, n=96 | -1.4 (9.34)
  Haemoglobin, Mon 24, n=110 | -2.2 (8.76)
  Haemoglobin, Mon 28, n=85 | -3.2 (9.49)
  Haemoglobin, Mon 32, n=86 | -2.2 (8.84)
  Haemoglobin, Mon 36, n=91 | -3.3 (10.04)
  Haemoglobin, Mon 40, n=78 | -3.4 (10.88)
  Haemoglobin, Mon 44, n=74 | -2.3 (9.74)
  Haemoglobin, Mon 48, n=79 | -4.3 (11.13)
  Haemoglobin, Mon 52, n=68 | -2.0 (9.51)
  Haemoglobin, Mon 56, n=63 | -2.8 (9.33)
  Haemoglobin, Mon 60, n=71 | -2.9 (10.15)
  Haemoglobin, Mon 64, n=49 | -3.7 (10.55)
  Haemoglobin, Mon 68, n=44 | -2.0 (10.41)
  Haemoglobin, Mon 72, n=53 | -3.8 (11.03)
  Haemoglobin, Mon 76, n=31 | -3.1 (11.65)
  Haemoglobin, Mon 80, n=24 | -3.7 (9.24)
  Haemoglobin, Mon 84, n=35 | -3.8 (11.97)
  Haemoglobin, Mon 88, n=16 | -3.1 (9.76)
  Haemoglobin, Mon 92, n=15 | 0.7 (9.14)
  Haemoglobin, Mon 96, n=19 | -2.1 (7.57)
  Haemoglobin, Mon 100, n=7 | 2.6 (8.87)
  Haemoglobin, Mon 104, n=1 | 8.0 (NA) — Standard deviation value was not available as only one participant was analyzed
  Haemoglobin, Mon 108, n=10 | 0.5 (7.47)

15. Primary Outcome: Change From Baseline in Chemistry Parameters-Alkaline Phosphatase (AP), Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST)
Description: Alkaline phosphatase (AP), Alanine aminotransferase (ALT), Aspartate aminotransferase (AST) were assessed at Month 1, Month 3, , Month 6, Month 9, Month 12 and every 4 months after Month 12. Baseline assessment in this study is defined as the last assessment for the endpoint in parent study taken prior to the first active treatment with Retigabine. Change from Baseline was calculated as post-Baseline value minus Baseline value. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles). NA indicates that data were not available.
Time Frame: Baseline and Up to Month 108
Population: Safety Population
Measure: Mean (Standard Deviation); unit: International units per litre (IU/L)
Arm/Group | Overall Study Arm
Number analyzed (Participants) | 181
International units per litre (IU/L)
  AP, Mon 1, n=151 | -5.5 (19.98)
  AP, Mon 3, n=136 | -5.7 (19.47)
  AP, Mon 6, n=122 | -7.3 (19.09)
  AP, Mon 9, n=108 | -7.7 (23.88)
  AP, Mon 12, n=149 | -6.1 (21.91)
  AP, Mon 16, n=87 | -9.1 (22.30)
  AP, Mon 20, n=85 | -5.0 (23.46)
  AP, Mon 24, n=95 | -7.1 (22.88)
  AP, Mon 28, n=75 | -6.3 (23.89)
  AP, Mon 32, n=73 | -7.8 (23.52)
  AP, Mon 36, n=77 | -4.8 (20.58)
  AP, Mon 40, n=67 | -6.3 (23.26)
  AP, Mon 44, n=63 | -8.2 (21.05)
  AP, Mon 48, n=70 | -7.5 (23.66)
  AP, Mon 52, n=59 | -9.7 (22.18)
  AP, Mon 56, n=54 | -9.9 (23.41)
  AP, Mon 60, n=61 | -7.7 (21.83)
  AP, Mon 64, n=44 | -2.8 (29.20)
  AP, Mon 68, n=36 | -8.7 (24.79)
  AP, Mon 72, n=46 | -4.5 (24.32)
  AP, Mon 76, n=26 | -5.0 (23.34)
  AP, Mon 80, n=21 | -8.9 (28.32)
  AP, Mon 84, n=30 | -1.7 (24.36)
  AP, Mon 88, n=15 | -9.9 (19.57)
  AP, Mon 92, n=15 | -6.5 (24.01)
  AP, Mon 96, n=18 | -3.9 (17.32)
  AP, Mon 100, n=6 | -12.3 (26.47)
  AP, Mon 104, n=1 | 11.0 (NA) — Standard deviation value was not available as only one participant was analyzed
  AP, Mon 108, n=9 | -14.2 (21.81)
  ALT, Mon 1, n=169 | 3.1 (16.74)
  ALT, Mon 3, n=152 | 4.0 (16.61)
  ALT, Mon 6, n=137 | 1.2 (10.45)
  ALT, Mon 9, n=122 | 5.2 (43.44)
  ALT, Mon 12, n=169 | 4.5 (26.42)
  ALT, Mon 16, n=100 | -0.3 (11.05)
  ALT, Mon 20, n=96 | 1.1 (10.89)
  ALT, Mon 24, n=108 | 3.0 (11.61)
  ALT, Mon 28, n=87 | 2.2 (12.65)
  ALT, Mon 32, n=85 | 2.0 (14.39)
  ALT, Mon 36, n=89 | 1.7 (10.36)
  ALT, Mon 40, n=77 | 2.5 (12.6)
  ALT, Mon 44, n=73 | 4.1 (13.29)
  ALT, Mon 48, n=78 | 3.0 (12.25)
  ALT, Mon 52, n=67 | 2.3 (12.15)
  ALT, Mon 56, n=62 | 1.4 (9.94)
  ALT, Mon 60, n=69 | 1.0 (11.73)
  ALT, Mon 64, n=48 | 0.2 (10.24)
  ALT, Mon 68, n=41 | -0.5 (9.11)
  ALT, Mon 72, n=51 | 0.4 (10.15)
  ALT, Mon 76, n=30 | 0.6 (6.14)
  ALT, Mon 80, n=22 | 0.4 (12.38)
  ALT, Mon 84, n=33 | 1.1 (12.05)
  ALT, Mon 88, n=15 | -1.3 (12.29)
  ALT, Mon 92, n=15 | 2.1 (8.09)
  ALT, Mon 96, n=18 | 2.2 (13.81)
  ALT, Mon 100, n=6 | 0.8 (9.41)
  ALT, Mon 104, n=1 | -6.0 (NA) — Standard deviation value was not available as only one participant was analyzed
  ALT, Mon 108, n=9 | -1.3 (6.86)
  AST, Mon 1, n=169 | 2.9 (10.79)
  AST, Mon 3, n=152 | 3.2 (10.07)
  AST, Mon 6, n=137 | 1.7 (7.89)
  AST, Mon 9, n=121 | 6.0 (35.18)
  AST, Mon 12, n=169 | 3.9 (14.84)
  AST, Mon 16, n=100 | 2.1 (8.49)
  AST, Mon 20, n=96 | 2.9 (8.03)
  AST, Mon 24, n=108 | 4.1 (9.72)
  AST, Mon 28, n=86 | 4.3 (9.16)
  AST, Mon 32, n=85 | 5.6 (8.64)
  AST, Mon 36, n=89 | 3.9 (6.74)
  AST, Mon 40, n=77 | 5.0 (9.93)
  AST, Mon 44, n=73 | 4.6 (7.84)
  AST, Mon 48, n=78 | 4.7 (8.61)
  AST, Mon 52, n=67 | 6.0 (8.68)
  AST, Mon 56, n=62 | 4.3 (7.61)
  AST, Mon 60, n=69 | 5.4 (9.34)
  AST, Mon 64, n=48 | 3.8 (8.50)
  AST, Mon 68, n=41 | 5.3 (7.13)
  AST, Mon 72, n=51 | 5.1 (9.54)
  AST, Mon 76, n=30 | 4.9 (6.59)
  AST, Mon 80, n=22 | 4.6 (7.74)
  AST, Mon 84, n=33 | 5.6 (8.60)
  AST, Mon 88, n=15 | 2.9 (6.99)
  AST, Mon 92, n=15 | 3.3 (3.24)
  AST, Mon 96, n=18 | 3.1 (6.58)
  AST, Mon 100, n=6 | 3.7 (4.23)
  AST, Mon 104, n=1 | 2.0 (NA) — Standard deviation value was not available as only one participant was analyzed
  AST, Mon 108, n=9 | 1.8 (5.49)

16. Primary Outcome: Change From Baseline in Chemistry Parameters-Bicarbonate, Blood Urea Nitrogen (BUN), Calcium, Chloride, Cholesterol, Non-fasting Glucose, Phosphorus, Potassium, Sodium, Urea
Description: Bicarbonate (Bic.), BUN, Calcium (Ca), Chloride (Cl), Cholesterol (Cho.), Non-fasting glucose (NFG), Phosphorus (P), Potassium (Ka), Sodium (Na), Urea were assessed at Month 1, Month 3, , Month 6, Month 9, Month 12 and every 4 months after Month 12. Baseline assessment in this study is defined as the last assessment for the endpoint in parent study taken prior to the first active treatment with Retigabine. Change from Baseline was calculated as post-Baseline value minus Baseline value. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles). NA indicates that data were not available.
Time Frame: Baseline and Up to Month 108
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimole per liter (mmol/L)
Arm/Group | Overall Study Arm
Number analyzed (Participants) | 181
Millimole per liter (mmol/L)
  BUN, Mon 3, n=142 | 0.843 (1.2012)
  BUN, Mon 6, n=130 | 0.917 (1.3506)
  BUN, Mon 9, n=115 | 0.823 (1.4786)
  BUN, Mon 12, n=156 | 0.717 (1.3707)
  BUN, Mon 16, n=94 | 0.973 (1.5385)
  BUN, Mon 20, n=92 | 1.060 (1.3001)
  BUN, Mon 24, n=102 | 0.809 (1.3654)
  BUN, Mon 28, n=82 | 0.876 (1.6420)
  BUN, Mon 32, n=80 | 0.942 (1.5201)
  BUN, Mon 36, n=85 | 0.958 (1.4267)
  BUN, Mon 40, n=72 | 1.135 (1.5626)
  BUN, Mon 44, n=69 | 0.844 (1.5006)
  BUN, Mon 48, n=75 | 0.952 (1.5679)
  BUN, Mon 52, n=62 | 1.071 (1.4554)
  BUN, Mon 56, n=57 | 1.022 (1.2697)
  BUN, Mon 60, n=64 | 1.100 (1.4931)
  BUN, Mon 64, n=44 | 0.991 (1.5938)
  BUN, Mon 68, n=37 | 1.148 (1.4599)
  BUN, Mon 72, n=48 | 1.087 (1.6218)
  BUN, Mon 76, n=27 | 1.257 (1.4492)
  BUN, Mon 80, n=19 | 0.939 (1.6115)
  BUN, Mon 84, n=30 | 0.929 (1.6810)
  BUN, Mon 88, n=15 | 0.881 (1.458)
  BUN, Mon 92, n=15 | 1.332 (1.9374)
  BUN, Mon 96, n=18 | 0.916 (1.8800)
  BUN, Mon 100, n=6 | 1.248 (1.5755)
  BUN, Mon 104, n=1 | 1.430 (NA) — Standard deviation value was not available as only one participant was analyzed
  BUN, Mon 108, n=9 | 0.183 (1.2637)
  Ca, Mon 1, n=170 | -0.034 (0.1094)
  Ca, Mon 3, n=152 | -0.013 (0.1107)
  Ca, Mon 6, n=137 | 0.012 (0.1035)
  Ca, Mon 9, n=123 | 0.020 (0.1006)
  Ca, Mon 12, n=169 | 0.024 (0.1167)
  Ca, Mon 16, n=100 | 0.042 (0.1143)
  Ca, Mon 20, n=97 | 0.052 (0.1180)
  Ca, Mon 24, n=109 | 0.049 (0.1095)
  Ca, Mon 28, n=87 | 0.034 (0.1135)
  Ca, Mon 32, n=85 | 0.032 (0.1216)
  Ca, Mon 36, n=89 | 0.032 (0.1176)
  Ca, Mon 40, n=77 | 0.030 (0.1195)
  Ca, Mon 44, n=73 | 0.040 (0.1093)
  Ca, Mon 48, n=80 | 0.054 (0.1161)
  Ca, Mon 52, n=67 | 0.047 (0.1170)
  Ca, Mon 56, n=62 | 0.055 (0.0951)
  Ca, Mon 60, n=69 | 0.061 (0.1184)
  Ca, Mon 64, n=49 | 0.056 (0.1338)
  Ca, Mon 68, n=41 | 0.083 (0.1245)
  Ca, Mon 72, n=51 | 0.053 (0.1223)
  Ca, Mon 76, n=30 | 0.097 (0.1341)
  Ca, Mon 80, n=22 | 0.069 (0.1289)
  Ca, Mon 84, n=34 | 0.106 (0.1023)
  Ca, Mon 88, n=15 | 0.071 (0.1078)
  Ca, Mon 92, n=15 | 0.116 (0.1013)
  Ca, Mon 96, n=18 | 0.106 (0.0887)
  Ca, Mon 100, n=6 | 0.148 (0.1217)
  Ca, Mon 104, n=1 | 0.170 (NA) — Standard deviation value was not available as only one participant was analyzed
  Ca, Mon 108, n=9 | 0.139 (0.1122)
  Cho., Mon 3, n=151 | 0.075 (0.6672)
  Cho., Mon 6, n=137 | 0.069 (0.6811)
  Cho., Mon 9, n=122 | 0.177 (0.7230)
  Cho., Mon 12, n=169 | 0.222 (0.7098)
  Cho., Mon 16, n=100 | 0.310 (0.7312)
  Cho., Mon 20, n=97 | 0.304 (0.7883)
  Cho., Mon 24, n=109 | 0.260 (0.7731)
  Cho., Mon 28, n=87 | 0.261 (0.7771)
  Cho., Mon 32, n=85 | 0.261 (0.8061)
  Cho., Mon 36, n=89 | 0.212 (0.8312)
  Cho., Mon 40, n=77 | 0.200 (0.7782)
  Cho., Mon 44, n=73 | 0.348 (0.7824)
  Cho., Mon 48, n=79 | 0.170 (0.8571)
  Cho., Mon 52, n=67 | 0.299 (0.7230)
  Cho., Mon 56, n=62 | 0.305 (0.7202)
  Cho., Mon 60, n=69 | 0.360 (0.7318)
  Cho., Mon 64, n=49 | 0.256 (0.8771)
  Cho., Mon 68, n=41 | 0.352 (0.8486)
  Cho., Mon 72, n=51 | 0.216 (0.8548)
  Cho., Mon 76, n=30 | 0.555 (0.7532)
  Cho., Mon 80, n=22 | 0.442 (0.7078)
  Cho., Mon 84, n=34 | 0.459 (0.9991)
  Cho., Mon 88, n=15 | 0.408 (0.7559)
  Cho., Mon 92, n=15 | 0.526 (0.7639)
  Cho., Mon 96, n=18 | 0.352 (0.628)
  Cho., Mon 100, n=6 | 0.483 (0.4126)
  Cho., Mon 104, n=1 | 0.160 (NA) — Standard deviation value was not available as only one participant was analyzed
  Cho., Mon 108, n=9 | 0.278 (0.3881)
  NFG, Mon 1, n=170 | 0.11 (0.929)
  NFG, Mon 3, n=149 | 0.20 (0.844)
  NFG, Mon 6, n=133 | 0.18 (1.057)
  NFG, Mon 9, n=120 | 0.38 (2.585)
  NFG, Mon 12, n=166 | 0.20 (0.978)
  NFG, Mon 16, n=100 | 0.18 (1.167)
  NFG, Mon 20, n=94 | 0.26 (0.971)
  NFG, Mon 24, n=106 | 0.13 (0.935)
  NFG, Mon 28, n=86 | 0.22 (0.968)
  NFG, Mon 32, n=85 | 0.16 (1.39)
  NFG, Mon 36, n=89 | 0.19 (1.176)
  NFG, Mon 40, n=75 | 0.20 (1.074)
  NFG, Mon 44, n=72 | 0.02 (1.019)
  NFG, Mon 48, n=77 | 0.27 (1.628)
  NFG, Mon 52, n=67 | 0.05 (0.877)
  NFG, Mon 56, n=61 | 0.14 (0.893)
  NFG, Mon 60, n=69 | 0.19 (1.029)
  NFG, Mon 64, n=49 | 0.21 (0.883)
  NFG, Mon 68, n=39 | 0.32 (0.700)
  NFG, Mon 72, n=51 | 0.24 (1.037)
  NFG, Mon 76, n=30 | 0.17 (0.505)
  NFG, Mon 80, n=22 | 0.15 (0.776)
  NFG, Mon 84, n=34 | 0.23 (0.572)
  NFG, Mon 88, n=15 | -0.09 (0.593)
  NFG, Mon 92, n=15 | 0.14 (0.546)
  NFG, Mon 96, n=18 | 0.22 (0.493)
  NFG, Mon 100, n=6 | 0.25 (0.176)
  NFG, Mon 104, n=1 | -0.50 (NA) — Standard deviation value was not available as only one participant was analyzed
  NFG, Mon 108, n=9 | 0.21 (0.372)
  P, Mon 1, n=169 | 0.014 (0.2037)
  P, Mon 3, n=148 | 0.001 (0.2029)
  P, Mon 6, n=132 | 0.020 (0.2148)
  P, Mon 9, n=119 | 0.021 (0.1974)
  P, Mon 12, n=167 | 0.007 (0.2401)
  P, Mon 16, n=100 | -0.010 (0.2289)
  P, Mon 20, n=94 | 0.003 (0.2229)
  P, Mon 24, n=105 | -0.021 (0.2186)
  P, Mon 28, n=86 | -0.020 (0.1974)
  P, Mon 32, n=84 | 0.019 (0.1767)
  P, Mon 36, n=88 | 0.004 (0.2896)
  P, Mon 40, n=75 | -0.005 (0.2408)
  P, Mon 44, n=73 | 0.018 (0.2631)
  P, Mon 48, n=78 | 0.019 (0.2165)
  P, Mon 52, n=67 | 0.018 (0.2160)
  P, Mon 56, n=62 | 0.010 (0.2330)
  P, Mon 60, n=69 | 0.071 (0.2389)
  P, Mon 64, n=49 | 0.027 (0.2722)
  P, Mon 68, n=39 | 0.007 (0.2453)
  P, Mon 72, n=51 | 0.029 (0.2761)
  P, Mon 76, n=30 | 0.038 (0.2506)
  P, Mon 80, n=22 | 0.107 (0.2761)
  P, Mon 84, n=34 | 0.046 (0.2518)
  P, Mon 88, n=15 | -0.004 (0.2970)
  P, Mon 92, n=15 | 0.058 (0.3334)
  P, Mon 96, n=18 | 0.026 (0.3294)
  P, Mon 100, n=6 | 0.143 (0.1656)
  P, Mon 104, n=1 | -0.090 (NA) — Standard deviation value was not available as only one participant was analyzed
  P, Mon 108, n=9 | -0.068 (0.3755)
  Ka, Mon 1, n=169 | 0.02 (0.416)
  Ka, Mon 3, n=149 | 0.04 (0.433)
  Ka, Mon 6, n=132 | 0.03 (0.362)
  Ka, Mon 9, n=119 | 0.08 (0.432)
  Ka, Mon 12, n=167 | -0.03 (0.442)
  Ka, Mon 16, n=100 | 0.02 (0.428)
  Ka, Mon 20, n=93 | 0.10 (0.442)
  Ka, Mon 24, n=106 | -0.00 (0.435)
  Ka, Mon 28, n=86 | -0.01 (0.437)
  Ka, Mon 32, n=84 | 0.01 (0.408)
  Ka, Mon 36, n=88 | 0.04 (0.482)
  Ka, Mon 40, n=74 | 0.00 (0.432)
  Ka, Mon 44, n=74 | 0.16 (0.538)
  Ka, Mon 48, n=79 | 0.12 (0.400)
  Ka, Mon 52, n=67 | 0.20 (0.448)
  Ka, Mon 56, n=62 | 0.08 (0.374)
  Ka, Mon 60, n=69 | 0.13 (0.511)
  Ka, Mon 64, n=49 | 0.19 (0.407)
  Ka, Mon 68, n=40 | 0.28 (0.394)
  Ka, Mon 72, n=52 | 0.24 (0.546)
  Ka, Mon 76, n=30 | 0.25 (0.549)
  Ka, Mon 80, n=22 | 0.35 (0.448)
  Ka, Mon 84, n=34 | 0.24 (0.483)
  Ka, Mon 88, n=15 | 0.38 (0.430)
  Ka, Mon 92, n=15 | 0.55 (0.503)
  Ka, Mon 96, n=18 | 0.41 (0.407)
  Ka, Mon 100, n=6 | 0.32 (0.402)
  Ka, Mon 104, n=1 | 1.10 (NA) — Standard deviation value was not available as only one participant was analyzed
  Ka, Mon 108, n=9 | 0.51 (0.437)
  Na, Mon 1, n=170 | 1.5 (3.44)
  Na, Mon 3, n=153 | 1.4 (2.88)
  Na, Mon 6, n=137 | 1.8 (3.16)
  Na, Mon 9, n=123 | 1.5 (3.22)
  Na, Mon 12, n=170 | 1.1 (3.68)
  Na, Mon 16, n=100 | 1.3 (3.26)
  Na, Mon 20, n=97 | 1.1 (3.33)
  Na, Mon 24, n=110 | 0.8 (3.57)
  Na, Mon 28, n=87 | 1.4 (3.06)
  Na, Mon 32, n=85 | 1.2 (3.46)
  Na, Mon 36, n=89 | 1.3 (3.84)
  Na, Mon 40, n=77 | 1.6 (3.78)
  Na, Mon 44, n=74 | 1.4 (3.78)
  Na, Mon 48, n=80 | 1.2 (3.31)
  Na, Mon 52, n=67 | 1.5 (4.09)
  Na, Mon 56, n=62 | 2.2 (3.21)
  Na, Mon 60, n=69 | 1.6 (3.46)
  Na, Mon 64, n=49 | 2.3 (3.63)
  Na, Mon 68, n=42 | 2.8 (3.64)
  Na, Mon 72, n=52 | 2.5 (3.60)
  Na, Mon 76, n=30 | 3.7 (3.43)
  Na, Mon 80, n=22 | 3.5 (4.15)
  Na, Mon 84, n=34 | 2.9 (4.04)
  Na, Mon 88, n=15 | 3.4 (3.18)
  Na, Mon 92, n=15 | 2.8 (2.46)
  Na, Mon 96, n=18 | 2.9 (2.24)
  Na, Mon 100, n=6 | 3.5 (4.09)
  Na, Mon 104, n=1 | 8.0 (NA) — Standard deviation value was not available as only one participant was analyzed
  Na, Mon 108, n=9 | 3.8 (4.35)
  Urea, Mon 1, n=13 | 0.712 (1.1012)
  Urea, Mon 3, n=10 | 0.533 (0.5127)
  Urea, Mon 6, n=7 | 0.304 (1.1204)
  Urea, Mon 9, n=8 | 0.846 (1.1121)
  Urea, Mon 12, n=13 | 0.713 (0.8743)
  Urea, Mon 16, n=6 | 1.070 (2.1793)
  Urea, Mon 20, n=5 | 0.856 (0.7814)
  Urea, Mon 24, n=8 | 0.668 (1.0143)
  Urea, Mon 28, n=5 | 1.498 (0.9608)
  Urea, Mon 32, n=5 | 0.784 (0.7722)
  Urea, Mon 36, n=4 | 1.337 (1.5564)
  Urea, Mon 40, n=5 | 1.140 (0.4659)
  Urea, Mon 44, n=5 | 0.784 (0.5269)
  Urea, Mon 48, n=5 | 0.712 (1.1305)
  Urea, Mon 52, n=5 | 0.356 (0.9411)
  Urea, Mon 56, n=5 | 1.356 (1.7009)
  Urea, Mon 60, n=5 | 1.282 (1.7228)
  Urea, Mon 64, n=5 | 1.496 (0.8128)
  Urea, Mon 68, n=4 | 1.695 (1.0242)
  Urea, Mon 72, n=3 | 1.070 (2.1725)
  Urea, Mon 76, n=3 | 1.070 (0.9430)
  Urea, Mon 80, n=3 | 2.380 (0.7398)
  Urea, Mon 84, n=4 | 1.695 (1.9006)
  Bicarbonate, Mon 1, n=169 | 0.4 (3.13)
  Bicarbonate, Mon 3, n=151 | 0.0 (3.27)
  Bicarbonate, Mon 6, n=136 | 0.4 (3.65)
  Bicarbonate, Mon 9, n=122 | 0.7 (3.48)
  Bicarbonate, Mon 12, n=169 | -0.0 (3.97)
  Bicarbonate, Mon 16, n=100 | 1.2 (3.49)
  Bicarbonate, Mon 20, n=97 | 1.5 (4.02)
  Bicarbonate, Mon 24, n=109 | 1.1 (3.28)
  Bicarbonate, Mon 28, n=87 | 1.6 (3.67)
  Bicarbonate, Mon 32, n=85 | 1.7 (3.62)
  Bicarbonate, Mon 36, n=89 | 1.6 (3.84)
  Bicarbonate, Mon 40, n=76 | 1.9 (3.89)
  Bicarbonate, Mon 44, n=73 | 2.7 (3.99)
  Bicarbonate, Mon 48, n=79 | 2.4 (3.43)
  Bicarbonate, Mon 52, n=66 | 2.8 (3.65)
  Bicarbonate, Mon 56, n=62 | 1.8 (3.79)
  Bicarbonate, Mon 60, n=69 | 2.4 (4.33)
  Bicarbonate, Mon 64, n=49 | 1.9 (3.95)
  Bicarbonate, Mon 68, n=42 | 2.0 (3.84)
  Bicarbonate, Mon 72, n=51 | 1.8 (3.59)
  Bicarbonate, Mon 76, n=30 | 2.2 (4.04)
  Bicarbonate, Mon 80, n=22 | 2.2 (3.74)
  Bicarbonate, Mon 84, n=34 | 3.0 (5.49)
  Bicarbonate, Mon 88, n=15 | 1.7 (2.09)
  Bicarbonate, Mon 92, n=15 | 1.7 (2.55)
  Bicarbonate, Mon 96, n=18 | 1.2 (3.73)
  Bicarbonate, Mon 100, n=6 | -0.7 (1.86)
  Bicarbonate, Mon 104, n=1 | 1.0 (NA) — Standard deviation value was not available as only one participant was analyzed
  Bicarbonate, Mon 108, n=9 | -0.4 (2.30)
  Cl, Mon 1, n=170 | 1.3 (3.38)
  Cl, Mon 3, n=153 | 1.3 (3.06)
  Cl, Mon 6, n=137 | 1.4 (3.32)
  Cl, Mon 9, n=123 | 1.6 (3.59)
  Cl, Mon 12, n=169 | 1.0 (3.73)
  Cl, Mon 16, n=100 | 1.8 (3.24)
  Cl, Mon 20, n=97 | 1.2 (3.56)
  Cl, Mon 24, n=110 | 1.0 (4.12)
  Cl, Mon 28, n=87 | 1.6 (3.45)
  Cl, Mon 32, n=85 | 1.8 (3.70)
  Cl, Mon 36, n=89 | 1.5 (4.00)
  Cl, Mon 40, n=77 | 1.6 (4.12)
  Cl, Mon 44, n=74 | 1.3 (3.81)
  Cl, Mon 48, n=80 | 1.2 (3.61)
  Cl, Mon 52, n=67 | 1.4 (4.13)
  Cl, Mon 56, n=61 | 2.0 (3.29)
  Cl, Mon 60, n=69 | 1.0 (3.77)
  Cl, Mon 64, n=49 | 1.7 (3.44)
  Cl, Mon 68, n=42 | 1.2 (3.62)
  Cl, Mon 72, n=52 | 1.6 (3.70)
  Cl, Mon 76, n=30 | 1.6 (4.11)
  Cl, Mon 80, n=22 | 2.0 (3.54)
  Cl, Mon 84, n=34 | 0.9 (3.53)
  Cl, Mon 88, n=15 | 2.2 (2.31)
  Cl, Mon 92, n=15 | 0.9 (3.11)
  Cl, Mon 96, n=18 | 0.7 (3.66)
  Cl, Mon 100, n=6 | 1.8 (4.26)
  Cl, Mon 104, n=1 | 1.0 (NA) — Standard deviation value was not available as only one participant was analyzed
  Cl, Mon 108, n=9 | 0.8 (3.56)

17. Primary Outcome: Change From Baseline in Chemistry Parameters -Creatinine, Total Bilirubin (TB), Uric Acid (UA)
Description: Creatinine, Total bilirubin (TB), Uric acid (UA) were assessed at Month 1, Month 3, , Month 6, Month 9, Month 12 and every 4 months after Month 12. Baseline assessment in this study is defined as the last assessment for the endpoint in parent study taken prior to the first active treatment with Retigabine. Change from Baseline was calculated as post-Baseline value minus Baseline value. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles). NA indicates that data were not available.
Time Frame: Baseline and Up to Month 108
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Micromole per Liter (umol/L)
Arm/Group | Overall Study Arm
Number analyzed (Participants) | 181
Micromole per Liter (umol/L)
  Creatinine, Mon 1, n=170 | 3 (12.20)
  Creatinine, Mon 3, n=149 | 4 (13.74)
  Creatinine, Mon 6, n=133 | 4.9 (13.47)
  Creatinine, Mon 9, n=120 | 3.7 (14.88)
  Creatinine, Mon 12, n=167 | 4.5 (13.91)
  Creatinine, Mon 16, n=100 | 4.0 (15.25)
  Creatinine, Mon 20, n=94 | 3.0 (15.67)
  Creatinine, Mon 24, n=105 | 1.9 (17.15)
  Creatinine, Mon 28, n=86 | -1.0 (13.98)
  Creatinine, Mon 32, n=84 | 0.0 (16.60)
  Creatinine, Mon 36, n=88 | -0.9 (14.90)
  Creatinine, Mon 40, n=75 | 0.1 (14.38)
  Creatinine, Mon 44, n=73 | -1.0 (13.93)
  Creatinine, Mon 48, n=79 | -0.2 (15.16)
  Creatinine, Mon 52, n=67 | 0.1 (14.84)
  Creatinine, Mon 56, n=62 | 1.2 (11.42)
  Creatinine, Mon 60, n=69 | -0.2 (15.54)
  Creatinine, Mon 64, n=49 | 0.6 (15.19)
  Creatinine, Mon 68, n=39 | 0.7 (14.31)
  Creatinine, Mon 72, n=51 | 0.1 (14.35)
  Creatinine, Mon 76, n=30 | 0.5 (14.75)
  Creatinine, Mon 80, n=22 | 3.3 (13.38)
  Creatinine, Mon 84, n=34 | 1.6 (18.72)
  Creatinine, Mon 88, n=15 | 1.2 (12.37)
  Creatinine, Mon 92, n=15 | 4.3 (12.45)
  Creatinine, Mon 96, n=18 | 1.2 (10.86)
  Creatinine, Mon 100, n=6 | 6.2 (12.06)
  Creatinine, Mon 104, n=1 | 9.0 (NA) — Standard deviation value was not available as only one participant was analyzed
  Creatinine, Mon 108, n=9 | 5.3 (14.40)
  TB Mon 1, n=167 | 4.6 (4.06)
  TB Mon 3, n=150 | 4.5 (4.34)
  TB Mon 6, n=134 | 3.8 (4.04)
  TB Mon 9, n=120 | 3.6 (4.40)
  TB Mon 12, n=167 | 2.7 (4.10)
  TB Mon 16, n=100 | 3.6 (4.41)
  TB Mon 20, n=97 | 3.7 (3.89)
  TB Mon 24, n=109 | 2.6 (4.10)
  TB Mon 28, n=87 | 2.8 (4.26)
  TB Mon 32, n=85 | 2.4 (4.95)
  TB Mon 36, n=89 | 2.2 (4.26)
  TB Mon 40, n=77 | 2.7 (4.68)
  TB Mon 44, n=73 | 2.6 (4.33)
  TB Mon 48, n=78 | 2.2 (4.98)
  TB Mon 52, n=67 | 2.0 (4.75)
  TB Mon 56, n=62 | 2.1 (4.54)
  TB Mon 60, n=68 | 2.1 (4.75)
  TB Mon 64, n=48 | 1.6 (4.56)
  TB Mon 68, n=41 | 1.2 (4.97)
  TB Mon 72, n=51 | 0.8 (4.64)
  TB Mon 76, n=29 | 1.0 (4.38)
  TB Mon 80, n=22 | 1.3 (3.69)
  TB Mon 84, n=34 | -0.3 (4.09)
  TB Mon 88, n=15 | 2.1 (7.05)
  TB Mon 92, n=15 | 1.3 (4.89)
  TB Mon 96, n=18 | -0.2 (5.06)
  TB Mon 100, n=6 | 1.2 (4.49)
  TB Mon 104, n=1 | 9.0 (NA) — Standard deviation value was not available as only one participant was analyzed
  TB Mon 108, n=9 | -0.3 (2.24)
  UA Mon 1, n=170 | 0.8 (39.49)
  UA Mon 3, n=152 | 3.1 (47.06)
  UA Mon 6, n=137 | 2.9 (44.98)
  UA Mon 9, n=123 | 4.5 (48.74)
  UA Mon 12, n=169 | 6.6 (50.88)
  UA Mon 16, n=100 | 2.5 (55.01)
  UA Mon 20, n=97 | 2.3 (49.72)
  UA Mon 24, n=109 | 4.7 (53.68)
  UA Mon 28, n=87 | 12.2 (51.73)
  UA Mon 32, n=85 | 10.2 (48.23)
  UA Mon 36, n=89 | 5.3 (52.19)
  UA Mon 40, n=77 | 6.9 (45.40)
  UA Mon 44, n=73 | 4.3 (53.75)
  UA Mon 48, n=79 | 5.7 (45.68)
  UA Mon 52, n=67 | 4.2 (52.86)
  UA Mon 56, n=62 | 8.6 (42.81)
  UA Mon 60, n=69 | 8.1 (49.74)
  UA Mon 64, n=49 | 2.7 (52.52)
  UA Mon 68, n=41 | 5.4 (52.49)
  UA Mon 72, n=51 | 12.6 (56.31)
  UA Mon 76, n=30 | 11.9 (53.61)
  UA Mon 80, n=22 | 7.0 (50.68)
  UA Mon 84, n=34 | 5.7 (58.19)
  UA Mon 88, n=15 | 3.1 (57.81)
  UA Mon 92, n=15 | -6.0 (60.45)
  UA Mon 96, n=18 | 5.3 (52.95)
  UA Mon 100, n=6 | 35.7 (62.78)
  UA Mon 104, n=1 | 107.0 (NA) — Standard deviation value was not available as only one participant was analyzed
  UA Mon 108, n=9 | 17.9 (59.95)

18. Primary Outcome: Change From Baseline in Chemistry Parameter-Total Protein
Description: Total Protein (TP) was assessed at Month 1, Month 3, , Month 6, Month 9, Month 12 and every 4 months after Month 12. Baseline assessment in this study is defined as the last assessment for the endpoint in parent study taken prior to the first active treatment with Retigabine. Change from Baseline was calculated as post-Baseline value minus Baseline value. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles)
Time Frame: Baseline and Up to Month 108
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Arm/Group | Overall Study
Number analyzed (Participants) | 181
Grams per liter (g/L)
  TP Mon 1, n=170 | -1.1 (4.44)
  TP Mon 3, n=152 | -0.5 (4.87)
  TP Mon 6, n=137 | -1.0 (4.77)
  TP Mon 9, n=123 | -0.8 (4.60)
  TP Mon 12, n=169 | 0.2 (4.45)
  TP Mon 16, n=100 | 0.3 (5.15)
  TP Mon 20, n=97 | 0.8 (4.64)
  TP Mon 24, n=109 | 0.2 (4.67)
  TP Mon 28, n=87 | -0.2 (4.52)
  TP Mon 32, n=85 | 0.1 (4.55)
  TP Mon 36, n=89 | -1.1 (4.48)
  TP Mon 40, n=77 | -1.1 (4.46)
  TP Mon 44, n=73 | -0.1 (4.72)
  TP Mon 48, n=79 | -1.3 (4.34)
  TP Mon 52, n=67 | -0.7 (4.67)
  TP Mon 56, n=62 | -1.1 (4.32)
  TP Mon 60, n=69 | -0.7 (4.75)
  TP Mon 64, n=49 | -0.2 (4.86)
  TP Mon 68, n=41 | 0.6 (4.82)
  TP Mon 72, n=51 | -0.7 (5.17)
  TP Mon 76, n=30 | 0.8 (4.93)
  TP Mon 80, n=22 | 0.3 (4.82)
  TP Mon 84, n=34 | 0.7 (5.90)
  TP Mon 88, n=15 | 0.4 (5.29)
  TP Mon 92, n=15 | 1.0 (4.09)
  TP Mon 96, n=18 | 0.9 (3.20)
  TP Mon 100, n=6 | 2.0 (4.77)
  TP Mon 104, n=1 | 7.0 (NA) — Standard deviation value was not available as only one participant was analyzed.
  TP Mon 108, n=9 | 2.1 (4.94)

19. Primary Outcome: Change From Baseline in Urine Specific Gravity
Description: Urine Specific gravity (USG) was assessed at Month 1, Month 3, , Month 6, Month 9, Month 12 and every 4 months after Month 12. Baseline assessment in this study is defined as the last assessment for the endpoint in parent study taken prior to the first active treatment with Retigabine. Change from Baseline was calculated as post-Baseline value minus Baseline value. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles). NA indicates that data were not available.
Time Frame: Baseline and Up to Month 108
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Dimensionless unit
Arm/Group | Overall Study
Number analyzed (Participants) | 181
Dimensionless unit
  USG, Mon 1, n=166 | -0.0018 (0.00848)
  USG, Mon 3, n=157 | -0.0016 (0.00852)
  USG, Mon 6, n=137 | 0.0002 (0.00930)
  USG, Mon 9, n=121 | 0.0002 (0.00933)
  USG, Mon 12, n=170 | -0.0000 (0.00937)
  USG, Mon 16, n=100 | 0.0006 (0.00960)
  USG, Mon 20, n=97 | 0.0008 (0.00964)
  USG, Mon 24, n=109 | -0.0012 (0.00985)
  USG, Mon 28, n=86 | -0.0003 (0.01032)
  USG, Mon 32, n=82 | -0.0006 (0.00935)
  USG, Mon 36, n=89 | -0.0024 (0.0086)
  USG, Mon 40, n=76 | -0.0005 (0.00865)
  USG, Mon 44, n=72 | -0.0007 (0.00867)
  USG, Mon 48, n=80 | -0.0015 (0.00941)
  USG, Mon 52, n=67 | 0.0002 (0.00972)
  USG, Mon 56, n=62 | -0.0003 (0.00899)
  USG, Mon 60, n=68 | -0.0023 (0.00893)
  USG, Mon 64, n=49 | -0.0022 (0.00938)
  USG, Mon 68, n=42 | -0.0022 (0.00822)
  USG, Mon 72, n=53 | -0.0015 (0.01006)
  USG, Mon 76, n=31 | -0.0024 (0.00822)
  USG, Mon 80, n=23 | -0.0021 (0.00867)
  USG, Mon 84, n=35 | -0.0028 (0.00862)
  USG, Mon 88, n=17 | -0.0055 (0.00833)
  USG, Mon 92, n=16 | -0.0030 (0.01116)
  USG, Mon 96, n=19 | -0.0039 (0.00956)
  USG, Mon 100, n=7 | -0.0013 (0.00886)
  USG, Mon 104, n=1 | -0.0150 (NA) — Standard deviation value was not available as only one participant was analyzed
  USG, Mon 108, n=10 | -0.0014 (0.01032)

20. Primary Outcome: Change From Baseline in Urine Power of Hydrogen (pH)
Description: Urine pH was assessed at Month 1, Month 3, , Month 6, Month 9, Month 12 and every 4 months after Month 12. Baseline assessment in this study is defined as the last assessment for the endpoint in parent study taken prior to the first active treatment with Retigabine. Change from Baseline was calculated as post-Baseline value minus Baseline value. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles). NA indicates that data were not available.
Time Frame: Baseline and Up to Month 108
Population: Safety Population
Measure: Mean (Standard Deviation); unit: pH units
Arm/Group | Overall Study
Number analyzed (Participants) | 181
pH units
  UpH, Mon 1, n=166 | -0.13 (0.721)
  UpH, Mon 3, n=157 | -0.18 (0.791)
  UpH, Mon 6, n=137 | -0.13 (0.767)
  UpH, Mon 9, n=121 | -0.17 (0.771)
  UpH, Mon 12, n=170 | -0.11 (0.793)
  UpH, Mon 16, n=100 | -0.05 (0.764)
  UpH, Mon 20, n=97 | -0.20 (0.886)
  UpH, Mon 24, n=109 | -0.09 (0.713)
  UpH, Mon 28, n=86 | -0.01 (0.893)
  UpH, Mon 32, n=82 | -0.10 (0.768)
  UpH, Mon 36, n=89 | 0.12 (0.83)
  UpH, Mon 40, n=76 | 0.09 (0.842)
  UpH, Mon 44, n=72 | 0.12 (0.767)
  UpH, Mon 48, n=80 | 0.19 (0.828)
  UpH, Mon 52, n=67 | 0.17 (0.851)
  UpH, Mon 56, n=62 | 0.06 (0.769)
  UpH, Mon 60, n=68 | 0.24 (0.896)
  UpH, Mon 64, n=49 | 0.19 (0.934)
  UpH, Mon 68, n=42 | 0.12 (0.825)
  UpH, Mon 72, n=53 | 0.16 (0.842)
  UpH, Mon 76, n=31 | 0.13 (1.000)
  UpH, Mon 80, n=23 | 0.24 (0.890)
  UpH, Mon 84, n=36 | 0.00 (0.862)
  UpH, Mon 88, n=17 | 0.21 (1.032)
  UpH, Mon 92, n=16 | 0.28 (1.224)
  UpH, Mon 96, n=19 | 0.26 (0.888)
  UpH, Mon 100, n=7 | 0.14 (1.180)
  UpH, Mon 104, n=1 | 0.50 (NA) — Standard deviation value was not available as only one participant was analyzed
  UpH, Mon 108, n=10 | 0.65 (0.747)

21. Primary Outcome: Change From Baseline in Post-void Residual Bladder Ultrasound Volume
Description: Post-void residual (PVR) bladder was assessed using ultrasound scan to assess urinary retention at Month 1, Month 3, Month 12 and annually after Month 12. Baseline assessment in this study is defined as the last assessment for the endpoint in parent study taken prior to the first active treatment with Retigabine. Change from Baseline was calculated as post-Baseline value minus Baseline value. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles)
Time Frame: Baseline and Up to Month 108
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Milliliter (mL)
Arm/Group | Overall Study
Number analyzed (Participants) | 181
Milliliter (mL)
  PVR, Mon 1, n=152 | 6.5 (60.92)
  PVR, Mon 3, n=146 | 5.8 (59.69)
  PVR, Mon 12, n=144 | -2.8 (73.95)
  PVR, Mon 24, n=75 | 11.6 (62.06)
  PVR, Mon 36, n=84 | 13.6 (58.45)
  PVR, Mon 48, n=77 | 8.8 (62.28)
  PVR, Mon 60, n=65 | 20.1 (85.81)
  PVR, Mon 72, n=48 | 17.2 (61.82)
  PVR, Mon 84, n=31 | 40.0 (89.38)
  PVR, Mon 96, n=19 | 8.7 (23.32)
  PVR, Mon 108, n=10 | 17.4 (60.89)

22. Primary Outcome: Change From Baseline in Overall American Urological Association (AUA) Symptom Index Score
Description: An AUA Symptom Index is a 7-item Likert-scored scale describing urinary bladder function and was completed by the Investigator to assess the participant's urinary voiding function at Month 1, Month 3, Month 12 and annually after Month 12. The index scale ranges from 0-35, where higher scores are indicative of a worse issue. Scores are categorized as 0-7 mild, 8-19 moderate and >19 severe. Baseline assessment in this study is defined as the last assessment for the endpoint in parent study taken prior to the first active treatment with Retigabine. Change from Baseline was calculated as post-Baseline value minus Baseline value. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles)
Time Frame: Baseline and Up to Month 108
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Overall Study
Number analyzed (Participants) | 181
Scores on a scale
  AUA, Mon 1, n=162 | -0.2 (6.17)
  AUA, Mon 3, n=151 | -0.0 (5.66)
  AUA, Mon 12, n=153 | 0.2 (6.30)
  AUA, Mon 24, n=79 | -0.1 (5.91)
  AUA, Mon 36, n=81 | 0.0 (4.62)
  AUA, Mon 48, n=79 | 0.5 (5.53)
  AUA, Mon 60, n=65 | 0.6 (4.42)
  AUA, Mon 72, n=49 | 0.4 (4.84)
  AUA, Mon 84, n=33 | 1.0 (4.89)
  AUA, Mon 96, n=19 | -1.0 (3.76)
  AUA, Mon 108, n=10 | -0.3 (5.06)

23. Primary Outcome: Number of Participants With Abnormal Results in Physical Examination
Description: A complete physical examination was performed at the end of each 12 month study cycle. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles). If a participant had an abnormal result for at least one body system of exam, that participant was included in the 'Abnormal' category
Time Frame: Up to Month 108
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Overall Study Arm
Number analyzed (Participants) | 181
Participants
  Baseline, n=181 | 59
  Mon 12, n=169 | 49
  Mon 24, n=113 | 34
  Mon 36, n=92 | 27
  Mon 48, n=82 | 25
  Mon 60, 69 | 32
  Mon 72, n=56 | 31
  Mon 84, n=36 | 25
  Mon 96, n=19 | 10
  Mon 108, n=10 | 5

24. Primary Outcome: Number of Participants With Abnormal Results of Neurological Examination
Description: Participants were assessed at Month 1, Month 3, Month 6, Month 9, Month 12 and every 4 months after Month 12. Participants in the worst category among the results of all neurological examination parameters are presented. Abnormal results were categorised as Abnormal not Clinically Significant (AbNCS)and Abnormal and Clinically Significant (AbCS). Only those participants available at the specified time points were analyzed (represented by n=X in the category titles)
Time Frame: Up to Month 108
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 181
Participants
  Baseline, n= 173, AbNCS | 60
  Baseline, n= 173, AbCS | 11
  Mon 1, n= 173, AbNCS | 49
  Mon 1, n= 173, AbCS | 17
  Mon 3, n= 159, AbNCS | 42
  Mon 3, n= 159, AbCS | 9
  Mon 6, n= 141, AbNCS | 35
  Mon 6, n= 141, AbCS | 8
  Mon 9, n= 125, AbNCS | 32
  Mon 9, n= 125, AbCS | 9
  Mon 12, n= 171, AbNCS | 56
  Mon 12, n= 171, AbCS | 13
  Mon 16, n= 104, AbNCS | 23
  Mon 16, n= 104, AbCS | 10
  Mon 20, n= 98, AbNCS | 28
  Mon 20, n= 98, AbCS | 6
  Mon 24, n= 113, AbNCS | 35
  Mon 24, n= 113, AbCS | 6
  Mon 28, n= 87, AbNCS | 23
  Mon 28, n= 87, AbCS | 6
  Mon 32, n= 86, AbNCS | 19
  Mon 32, n= 86, AbCS | 5
  Mon 36, n= 92, AbNCS | 28
  Mon 36, n= 92, AbCS | 6
  Mon 40, n= 78, AbNCS | 22
  Mon 40, n= 78, AbCS | 8
  Mon 44, n= 76, AbNCS | 25
  Mon 44, n= 76, AbCS | 3
  Mon 48, n= 82, AbNCS | 25
  Mon 48, n= 82, AbCS | 6
  Mon 52, n= 67, AbNCS | 19
  Mon 52, n= 67, AbCS | 4
  Mon 56, n= 63, AbNCS | 19
  Mon 56, n= 63, AbCS | 4
  Mon 60, n= 68, AbNCS | 27
  Mon 60, n= 68, AbCS | 3
  Mon 64, n= 50, AbNCS | 21
  Mon 64, n= 50, AbCS | 1
  Mon 68, n= 44, AbNCS | 15
  Mon 68, n= 44, AbCS | 0
  Mon 72, n= 56, AbNCS | 20
  Mon 72, n= 56, AbCS | 4
  Mon 76, n= 31, AbNCS | 11
  Mon 76, n= 31, AbCS | 0
  Mon 80, n= 24, AbNCS | 7
  Mon 80, n= 24, AbCS | 0
  Mon 84, n= 36, AbNCS | 14
  Mon 84, n= 36, AbCS | 0
  Mon 88, n= 17, AbNCS | 0
  Mon 88, n= 17, AbCS | 1
  Mon 92, n= 16, AbNCS | 2
  Mon 92, n= 16, AbCS | 1
  Mon 96, n= 19, AbNCS | 4
  Mon 96, n= 19, AbCS | 0
  Mon 100, n= 7, AbNCS | 2
  Mon 100, n= 7, AbCS | 0
  Mon 104, n= 1, AbNCS | 1
  Mon 104, n= 1, AbCS | 0
  Mon 108, n= 10, AbNCS | 2
  Mon 108, n= 10, AbCS | 0

25. Primary Outcome: Number of Participants With Pigmentation of Non-retinal Ocular Tissue
Description: The ophthalmologist/retina specialist determined the presence or absence of abnormal discoloration of all non-retinal ocular tissues. Only those participants available at the specified time points were analyzed.
Time Frame: Assessed up to a maximum of 9 years
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 36
Participants | 11

26. Primary Outcome: Number of Participants With Pigmentation of Retinal Ocular Tissue
Description: The ophthalmologist/retina specialist determined the presence or absence of abnormal discoloration of retinal ocular tissues. It included Pigmentary abnormalities in the macula, of peripheral retina as well as in both of them.. Only those participants available at the specified time points were analyzed.
Time Frame: Assessed up to a maximum of 9 years
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 36
Participants | 14

27. Primary Outcome: Number of Participants With Abnormal Pigmentation of Skin, Including the Skin Around the Eyes and the Eyelids, Lips, Nails, or Mucosa
Description: An assessment of the participant's nails, lips, skin and mucosa was completed by the investigator at the 4 monthly study visits. The assessment of the participant's skin included assessment of the skin around the eyes and the eyelids,lips, nails, and mucosa
Time Frame: Assessed up to a maximum of 9 years
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 181
Participants
  Any abnormal dermatologic discoloration | 23
  Abnormal discoloration of skin | 15
  Abnormal discoloration of lips | 16
  Abnormal discoloration of nails | 21
  Abnormal discoloration of mucosa | 17
  Abnormal discoloration of sun-exposed tissue | 22
  Abnormal discoloration of non su-exposed tissue | 18

28. Primary Outcome: Number of Participants With a Clinically Significant Decrease in Visual Acuity From Initial Examination
Description: A comprehensive eye examination was conducted by retina specialist or general ophthalmologist to assess best corrected visual acuity. An initial comprehensive eye examination was completed by an ophthalmologist for all participants. This exam was not associated with a specific visit. Thereafter, eye examinations was performed approximately every 6 months. Eye examination was introduced following protocol amendment and was conducted in all participants. Participants discontinued before implementation of this amendment and who have not had a comprehensive eye examination and skin examination (and follow-up by a dermatologist, if clinically indicated) were asked to return to the clinic for an evaluation of their skin (and follow-up dermatology examination, if clinically indicated) and for a comprehensive eye examination. Number of Par. with both initial and at least one follow-up exam while on RTG treatment were analyzed.
Time Frame: Assessed up to a maximum of 9 years
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 24
Participants | 2

29. Primary Outcome: Number of Participants With a Decrease in Confrontational Visual Field From Initial Examination
Description: Decrease in confrontation visual field is defined as a participant having a normal initial exam and an abnormal exam thereafter or, a response of clinically significant worsening in either eye since the last assessment.
Time Frame: Assessed up to a maximum of 9 years
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 181
Participants | 0

30. Primary Outcome: Number of Participants With Resolution of Abnormal Eye Pigmentation After Discontinuation of Retigabine
Description: The ophthalmologist/retina specialist determined the presence or absence of retinal and non-retinal ocular abnormalities. Retinal abnormalities included abnormalities in the macula and/or the peripheral retina and non-retinal ocular pigmentary abnormality.
Time Frame: 2 years and 9 months
Population: All SFUCP Subjects Population included participants with one or more finding(s) of abnormal pigmentation of the retina or unexplained vision loss, pigmentation of non-retinal ocular tissue or discoloration of skin, lips, nails or mucosa at the treatment phase withdrawal/follow-up visit and who enter the SFUCP phase.
Measure: Number; unit: Participants
Groups:
- Retigabine SFUCP: Participants who withdraw from retigabine and who were found to have abnormal pigmentation of the retina or unexplained vision loss, pigmentation of non-retinal ocular tissue or discoloration of skin, lips, nails or mucosa entered the SFUCP. During the SFUCP, participants underwent 6-monthly comprehensive eye examinations and/or skin assessments by the investigator, ophthalmologist, retinal specialist or dermatologist as appropriate. Participants were followed up in the SFUCP until the dermatology/ophthalmology finding(s) either resolved or stabilized. Stabilization was defined in the protocol as no changes on two consecutive 6-monthly assessments over at least over 12 months after discontinuation of retigabine.
Arm/Group | Retigabine SFUCP
Number analyzed (Participants) | 19
Participants
  Retinal pigmentary abnormality | 1
  Pigmentary abnormality of macula | 1
  Pigmentary abnormality of peripheral retina | 3
  Non-retinal ocular pigmentary abnormality | 4

31. Primary Outcome: Number of Participants With Resolution of Dermatologist Confirmed Abnormal Discoloration After Discontinuation of Retigabine
Description: An assessment of the participant's nails, lips, skin and mucosa was completed by the investigator at the 6 monthly SFUCP study visits. The assessment of the participant's skin included assessment of the skin around the eyes and the eyelids, lips, nails, and mucosa.
Time Frame: 2 years 9 months
Population: All SFUCP Subjects Population
Measure: Number; unit: Participants
Arm/Group | Retigabine SFUCP
Number analyzed (Participants) | 19
Participants | 1

32. Primary Outcome: Time From Discontinuation of Retigabine to Resolution of Abnormal Eye Pigmentation
Description: Retinal pigmentary abnormality was determined by either an ophthalmologist or retina specialist. Retinal pigmentary abnormality included pigmentary abnormality of macula, pigmentary abnormality of the peripheral retina and non-retinal ocular pigmentary abnormality. If a participant had pigmentary abnormality of macula and pigmentary abnormality of the peripheral retina both should be resolved in order for retinal pigmentary abnormality to be considered resolved. If a participant had non-retinal ocular pigmentary abnormality in more than location (conjunctiva, sclera, cornea, iris or lens), all should be resolved for non-retinal pigmentary abnormality to be considered resolved. Only participants with resolution of the specified pigmentation are included in this analysis.
Time Frame: 2 years 9 months
Population: All SFUCP Subjects Population
Measure: Median (Full Range); unit: Days
Arm/Group | Retigabine SFUCP
Number analyzed (Participants) | 19
Days
  Retinal Pigmentary Abnormality, n=1: number analyzed (Participants) | 1
  Retinal Pigmentary Abnormality, n=1 | 317.0 [317 to 317]
  Pigmentary Abnormality of Macula, n=1: number analyzed (Participants) | 1
  Pigmentary Abnormality of Macula, n=1 | 163.0 [163 to 163]
  Pigmentary Abnormality of Peripheral Retina, n=3: number analyzed (Participants) | 3
  Pigmentary Abnormality of Peripheral Retina, n=3 | 317.0 [197 to 794]
  Non-Retinal Ocular Pigmentary Abnormality, n=4: number analyzed (Participants) | 4
  Non-Retinal Ocular Pigmentary Abnormality, n=4 | 180.0 [34 to 561]

33. Primary Outcome: Time From Discontinuation of Retigabine to Resolution of All Dermatologist-Confirmed Abnormal Discoloration
Description: Assessments were at approximately 6-monthly intervals (timed relative to the participants previous dermatology assessment) until the abnormal discoloration either resolved or stabilized (as defined by no changes over 2 consecutive 6-monthly assessments performed by the dermatologist over at least 12 months after discontinuation of retigabine). The assessment of the participant's skin included assessment of the skin around the eyes and the eyelids, lips, nails, and mucosa. Only participants with resolution of the specified tissue are included in this analysis.
Time Frame: 2 years 9 months
Population: All SFUCP Subjects Population
Measure: Median (Full Range); unit: Days
Arm/Group | Retigabine SFUCP
Number analyzed (Participants) | 19
Days
  All, n=1: number analyzed (Participants) | 1
  All, n=1 | 439.0 [439 to 439]
  Skin, n=5: number analyzed (Participants) | 5
  Skin, n=5 | 347.0 [203 to 952]
  Lips, n=4: number analyzed (Participants) | 4
  Lips, n=4 | 284.5 [133 to 590]
  Nails,n=7: number analyzed (Participants) | 7
  Nails,n=7 | 377.0 [203 to 762]
  Mucosa, n=3: number analyzed (Participants) | 3
  Mucosa, n=3 | 468.0 [133 to 541]

34. Secondary Outcome: Percentage Change From Baseline in the 28-day Partial Seizure
Description: Twenty-eight-day total partial seizure frequency during the study is defined as the sum of total partial seizures from First date (Baseline visit date +1 if no seizures on Baseline or Baseline visit date if seizures reported on the Baseline) to Last date (last visit date for seizure record with non-missing response), divided by applicable days, standardized by 28 days. The applicable days are the days in which the subject had non-missing seizure data. Change from Baseline was calculated as post-Baseline value minus Baseline value. Only those participants available at the specified time points were analyzed.
Time Frame: Assessed up to a maximum of 9 years
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Overall Study
Number analyzed (Participants) | 179
Percent change | -34.2 (68.70)

35. Secondary Outcome: Number of Responders
Description: A participant was classified as a responder if there is an at least 50% reduction from Baseline in the 28-day total Partial Seizure frequency. Baseline was defined as the parent study Baseline. Only those participants available at the specified time points were analyzed.
Time Frame: Assessed up to a maximum of 9 years
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 179
Participants | 98

36. Secondary Outcome: Number of Participants Who Were Seizure Free for Any 6 Continuous Months
Description: Number of seizure free days is defined as the number of applicable days without any seizures (partial, generalized or unclassified). Only the days in which a subject had non-missing seizure data were considered as applicable days. Duration of exposure is defined using a window range allowed for each scheduled visit. At least 6 months of exposure is defined as >= 173 days of exposure since the window range for Month 6 visit is +/- 7 days. Only those participants available at the specified time points were analyzed.
Time Frame: Assessed up to a maximum of 9 years
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 140
Participants | 20

37. Secondary Outcome: Number of Participants Who Were Seizure Free for Any 12 Continuous Months
Description: Duration of exposure is defined using a window range allowed for each scheduled visit. At least 12 months of exposure is defined as >= 353 days of exposure since the window range for Month 12 visit is +/- 7 days. Only those participants available at the specified time points were analyzed.
Time Frame: Assessed up to a maximum of 9 years
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 112
Participants | 14

38. Secondary Outcome: Percentage of Seizure-free Days
Description: Number of seizure free days is defined as the number of applicable days without any seizures (partial, generalized or unclassified). Only the days in which a participant had non-missing seizure data was considered as applicable days
Time Frame: Assessed up to a maximum of 9 years
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Percentage of days
Arm/Group | Overall Study
Number analyzed (Participants) | 179
Percentage of days | 75.7 (25.92)

39. Secondary Outcome: Change From Baseline in Quality of Life in Epilepsy (QOLIE)-31-P Questionnaire
Description: The QOLIE-31-P (Version 2.0) was utilized to assess quality of life. The QOLIE-31-P assessment was completed by the participants at Baseline, Month 3, Month 6, Month 9, Month 12 and annually after Month 12. The QOLIE has 7 sub scales as energy fatigue, emotional well being, social functioning, cognitive, medication effects, seizure worry and overall QOL. The assessment range for the overall score and the sub-scales is 0-100, where higher scores indicate greater well being. Change from Baseline was calculated as post-Baseline value minus Baseline value. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles)
Time Frame: Assessed up to a maximum of 9 years
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Overall Study
Number analyzed (Participants) | 181
Scores on a scale
  Mon 3, n= 133 | -2 (12.992)
  Mon 6, n= 130 | -2.95 (12.729)
  Mon 9, n= 114 | -1.65 (13.074)
  Mon 12, n= 156 | -2.77 (13.616)
  Mon 24, n= 102 | -3.13 (13.602)
  Mon 36, n= 81 | -2.43 (13.925)
  Mon 48, n= 74 | -1.05 (12.605)
  Mon 60, n= 60 | -0.41 (13.309)
  Mon 72, n= 49 | -0.35 (14.382)
  Mon 84, n= 28 | 0.19 (14.699)
  Mon 96, n= 18 | -0.25 (17.986)
  Mon 108, n= 11 | 1.55 (18.768)

ADVERSE EVENTS:
Time Frame: SAEs and non-serious AEs were collected from 1st dose of study medication in the OLE until 30 days after stopping study drug. Any AEs from parent study that worsened during the OLE are also captured (Assessed up to a maximum of 9 years).
Description: SAEs and non-serious AEs were assessed in the Safety Population
Arm/Group | Overall Study
All-Cause Mortality (participants affected / at risk) | 1/181
Serious Adverse Events (participants affected / at risk) | 48/181
Other Adverse Events (participants affected / at risk) | 169/181
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Overall Study (N=181)
Toxicity to various agents (Injury, poisoning and procedural complications) | 2
Ankle fracture (Injury, poisoning and procedural complications) | 1
Burns second degree (Injury, poisoning and procedural complications) | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 1
Hand fracture (Injury, poisoning and procedural complications) | 1
Head injury (Injury, poisoning and procedural complications) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Jaw fracture (Injury, poisoning and procedural complications) | 1
Joint injury (Injury, poisoning and procedural complications) | 1
Laceration (Injury, poisoning and procedural complications) | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 1
Radius fracture (Injury, poisoning and procedural complications) | 1
Splenic injury (Injury, poisoning and procedural complications) | 1
Seizure (Nervous system disorders) | 4
Epilepsy (Nervous system disorders) | 2
Cerebrovascular accident (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Hemiparesis (Nervous system disorders) | 1
Lumbar radiculopathy (Nervous system disorders) | 1
Partial seizures with secondary generalisation (Nervous system disorders) | 1
Postictal state (Nervous system disorders) | 1
Psychomotor hyperactivity (Nervous system disorders) | 1
Seizure cluster (Nervous system disorders) | 1
Status epilepticus (Nervous system disorders) | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1
Tonic convulsion (Nervous system disorders) | 1
Pneumonia (Infections and infestations) | 6
Urinary tract infection (Infections and infestations) | 3
Anal abscess (Infections and infestations) | 1
Appendicitis perforated (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Confusional state (Psychiatric disorders) | 1
Conversion disorder (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Epileptic psychosis (Psychiatric disorders) | 1
Major depression (Psychiatric disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Nervousness (Psychiatric disorders) | 1
Somatic Symptom Disorder (Psychiatric disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 2
Abdominal adhesions (Gastrointestinal disorders) | 1
Neutropenic Colitis (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Insulinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bile duct obstruction (Hepatobiliary disorders) | 1
Biliary colic (Hepatobiliary disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Clostridium test positive (Investigations) | 1
Liver function test abnormal (Investigations) | 1
Transaminases increased (Investigations) | 1
Urinary retention (Renal and urinary disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Angina unstable (Cardiac disorders) | 1
Idiosyncratic drug reaction (General disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Overall Study (N=181)
Dizziness (Nervous system disorders) | 55
Somnolence (Nervous system disorders) | 44
Headache (Nervous system disorders) | 42
Urinary tract infection (Renal and urinary disorders) | 37
Influenza (Infections and infestations) | 28
Tremor (Nervous system disorders) | 22
Oral mucosal discolouration (Gastrointestinal disorders) | 21
Fatigue (General disorders) | 20
Seizure (Nervous system disorders) | 16
Skin discolouration (Skin and subcutaneous tissue disorders) | 19
Abdominal pain (Gastrointestinal disorders) | 18
Back pain (Musculoskeletal and connective tissue disorders) | 18
Contusion (Injury, poisoning and procedural complications) | 17
Dysarthria (Nervous system disorders) | 17
Paraesthesia (Nervous system disorders) | 17
Diarrhoea (Gastrointestinal disorders) | 16
Lip discolouration (Gastrointestinal disorders) | 16
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 16
Nail discolouration (Skin and subcutaneous tissue disorders) | 15
Nail pigmentation (Skin and subcutaneous tissue disorders) | 15
Pigmentation lip (Gastrointestinal disorders) | 15
Vomiting (Gastrointestinal disorders) | 15
Anxiety (Psychiatric disorders) | 14
Constipation (Gastrointestinal disorders) | 14
Nausea (Gastrointestinal disorders) | 14
Depression (Psychiatric disorders) | 13
Memory impairment (Nervous system disorders) | 13
Viral Upper Respiratory Tract Infection (Infections and infestations) | 10
Toothache (Gastrointestinal disorders) | 13
Urinary retention (Renal and urinary disorders) | 11
Ataxia (Nervous system disorders) | 12
Laceration (Injury, poisoning and procedural complications) | 11
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12
Sinusitis (Infections and infestations) | 12
Amnesia (Nervous system disorders) | 11
Aphasia (Nervous system disorders) | 11
Retinal pigmentation (Eye disorders) | 11
Vertigo (Ear and labyrinth disorders) | 11
Vision blurred (Eye disorders) | 11
Abdominal pain upper (Gastrointestinal disorders) | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 10
Diplopia (Eye disorders) | 10
Speech disorder (Nervous system disorders) | 10
Urinary hesitation (Renal and urinary disorders) | 10
Confusional state (Psychiatric disorders) | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.